CLINICAL TRIAL: NCT01871805
Title: A Phase I/II Study of the ALK Inhibitor CH5424802/ RO5424802 in Patients With ALK-Rearranged Non-Small Cell Lung Cancer Previously Treated With Crizotinib
Brief Title: A Study of Alectinib (CH5424802/RO5424802) in Participants With Anaplastic Lymphoma Kinase (ALK)-Rearranged Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP28761; NCT01588028 (obsolete NCT alias)
Record Dates: First submitted 2013-05-28; First posted 2013-06-07 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib

ARMS (2):
- Alectinib: Phase I (Dose Escalation) (Experimental): Participants will receive escalating doses of alectinib capsules orally until disease progression, death or withdrawal for any other reasons.
  Interventions: Drug: Alectinib
- Alectinib (Phase II: RP2 dose) (Experimental): Participants will receive recommended Phase II dose as determined from Phase I until disease progression, death or withdrawal for any other reasons.
  Interventions: Drug: Alectinib

INTERVENTIONS:
Drug: Alectinib — Participants will receive alectinib as described in the arm descriptions.
  Other Names: CH5424802; RO5424802

SUMMARY:
This non-randomized, open-label, multicenter study will evaluate the safety and efficacy of alectinib in participants with ALK-rearranged non-small cell lung cancer who failed crizotinib treatment. In Phase I, cohorts of participants will receive escalating doses of alectinib orally twice daily. In Phase II, patients who failed crizotinib treatment will receive the recommended phase II dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, locally advanced, not amenable to curative therapy, or metastatic NSCLC
* ALK-rearrangement confirmed by the Food and Drug Administration (FDA) approved test
* NSCLC that has failed crizotinib treatment
* Measurable disease as defined by RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to (<=) 2
* Adequate hematologic, hepatic and renal function

Exclusion Criteria:

* Prior therapy with ALK inhibitor other than crizotinib
* Brain or leptomeningeal metastases that are symptomatic and/or requiring treatment
* History of serious cardiac dysfunction
* History of or current active infection with hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
* Clinically significant gastrointestinal abnormality that would affect absorption of the drug
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2014-10-24 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (42):
- United States (39):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Irvine, Irvine, California
  - UCSD Moores Cancer Center, La Jolla, California
  - Loma Linda Cancer Center, Loma Linda, California
  - UCLA, Los Angeles, California
  - Univ of Colorado Canc Ctr, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Lynn Regional Cancer Center West, Boca Raton, Florida
  - Florida Hospital Cancer Inst, Orlando, Florida
  - UF Health Orlando, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Inst., Tampa, Florida
  - University of Illinois Cancer Center, Chicago, Illinois
  - Monroe Medical Associates; Ingalls Memorial Hosp, Harvey, Illinois
  - Massachussets General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Can Ins, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - St. Joseph Mercy Hospital; Cancer Care Center., Ann Arbor, Michigan
  - Wayne State Uni ; Karmanos Cancer Center, Detroit, Michigan
  - Hackensack Univ Med Ctr, Hackensack, New Jersey
  - Roswell Park Cancer Inst., Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, Commack, New York
  - Richmond University Medical Center; Pharmacy Department, Staten Island, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Providence Portland Med Ctr, Portland, Oregon
  - Oregon Health & Science Uni, Portland, Oregon
  - St. Luke's Hospital; Pharmacy Department, Bethlehem, Pennsylvania
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Pavillion, Pittsburgh, Pennsylvania
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - Center for Biomedical Research LLC, Knoxville, Tennessee
  - Texas Oncology-Baylor Sammons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Swedish Cancer Inst., Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Lakeridge Health Oshawa; Oncology, Oshawa, Ontario
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec

REFERENCES:
- [Derived] Gadgeel S, Shaw AT, Barlesi F, Crino L, Yang JC, Dingemans AM, Kim DW, de Marinis F, Schulz M, Liu S, Gupta R, Smoljanovic V, Ou SI. Time To Response In Patients With Advanced Anaplastic Lymphoma Kinase (ALK)-Positive Non-Small-Cell Lung Cancer (NSCLC) Receiving Alectinib In The Phase II NP28673 And NP28761 Studies. Lung Cancer (Auckl). 2019 Nov 13;10:125-130. doi: 10.2147/LCTT.S209231. eCollection 2019. PMID 32009824
- [Derived] Ou SI, Gadgeel SM, Barlesi F, Yang JC, De Petris L, Kim DW, Govindan R, Dingemans AM, Crino L, Lena H, Popat S, Ahn JS, Dansin E, Mitry E, Muller B, Bordogna W, Balas B, Morcos PN, Shaw AT. Pooled overall survival and safety data from the pivotal phase II studies (NP28673 and NP28761) of alectinib in ALK-positive non-small-cell lung cancer. Lung Cancer. 2020 Jan;139:22-27. doi: 10.1016/j.lungcan.2019.10.015. Epub 2019 Oct 14. PMID 31706099
- [Derived] Morcos PN, Nueesch E, Jaminion F, Guerini E, Hsu JC, Bordogna W, Balas B, Mercier F. Exposure-response analysis of alectinib in crizotinib-resistant ALK-positive non-small cell lung cancer. Cancer Chemother Pharmacol. 2018 Jul;82(1):129-138. doi: 10.1007/s00280-018-3597-5. Epub 2018 May 10. PMID 29748847
- [Derived] Gadgeel SM, Shaw AT, Govindan R, Gandhi L, Socinski MA, Camidge DR, De Petris L, Kim DW, Chiappori A, Moro-Sibilot DL, Duruisseaux M, Crino L, De Pas T, Dansin E, Tessmer A, Yang JC, Han JY, Bordogna W, Golding S, Zeaiter A, Ou SI. Pooled Analysis of CNS Response to Alectinib in Two Studies of Pretreated Patients With ALK-Positive Non-Small-Cell Lung Cancer. J Clin Oncol. 2016 Dec;34(34):4079-4085. doi: 10.1200/JCO.2016.68.4639. Epub 2016 Oct 31. PMID 27863201
- [Derived] Lin YT, Yu CJ, Yang JC, Shih JY. Anaplastic Lymphoma Kinase (ALK) Kinase Domain Mutation Following ALK Inhibitor(s) Failure in Advanced ALK Positive Non-Small-Cell Lung Cancer: Analysis and Literature Review. Clin Lung Cancer. 2016 Sep;17(5):e77-e94. doi: 10.1016/j.cllc.2016.03.005. Epub 2016 Mar 30. PMID 27130468
- [Derived] Shaw AT, Gandhi L, Gadgeel S, Riely GJ, Cetnar J, West H, Camidge DR, Socinski MA, Chiappori A, Mekhail T, Chao BH, Borghaei H, Gold KA, Zeaiter A, Bordogna W, Balas B, Puig O, Henschel V, Ou SI; study investigators. Alectinib in ALK-positive, crizotinib-resistant, non-small-cell lung cancer: a single-group, multicentre, phase 2 trial. Lancet Oncol. 2016 Feb;17(2):234-242. doi: 10.1016/S1470-2045(15)00488-X. Epub 2015 Dec 19. Erratum In: Lancet Oncol. 2017 Mar;18(3):e134. doi: 10.1016/S1470-2045(17)30077-3. PMID 26708155
- [Derived] Gadgeel SM, Gandhi L, Riely GJ, Chiappori AA, West HL, Azada MC, Morcos PN, Lee RM, Garcia L, Yu L, Boisserie F, Di Laurenzio L, Golding S, Sato J, Yokoyama S, Tanaka T, Ou SH. Safety and activity of alectinib against systemic disease and brain metastases in patients with crizotinib-resistant ALK-rearranged non-small-cell lung cancer (AF-002JG): results from the dose-finding portion of a phase 1/2 study. Lancet Oncol. 2014 Sep;15(10):1119-28. doi: 10.1016/S1470-2045(14)70362-6. Epub 2014 Aug 18. PMID 25153538

RESULTS

PARTICIPANT FLOW:
Groups:
- Alectinib 300 mg (Fasted): Phase I: Participants received single dose of 20 or 40 milligrams (mg) alectinib capsules orally to make a dose of 240 or 300 mg on Cycle 1 Day -3 and then received 300 mg twice daily (BID) dose for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
- Alectinib 460 mg (Fed): Phase I: Participants received single dose of 20 or 40 mg alectinib capsules orally to make a dose of 460 mg on Cycle 1 Day -3 and then received 460 mg BID dose for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
- Alectinib 600 mg (Fed): Phase I (20/40/150 mg): Participants received single dose of 20 or 40 or 150 mg alectinib capsules orally to make a dose of 600 mg on Cycle 1 Day -3 and then received 600 mg BID dose for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
- Alectinib 760 mg (Fed): Phase I: Participants received single dose of 20 or 40 mg alectinib capsules orally to make a dose of 760 mg on Cycle 1 Day -3 and then received 760 mg BID dose for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
- Alectinib 900 mg (Fed): Phase I (20/40/150 mg): Participants received single dose of 20 or 40 or 150 mg alectinib capsules orally to make a dose of 900 mg on Cycle 1 Day -3 and then received 900 mg BID dose for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
- Alectinib 600 mg (Fed): Phase II: Participants received 150 mg alectinib capsules orally to make a dose of 600 mg BID from Cycle 1 Day 1 for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
Period: Phase I
Arm/Group | Alectinib 300 mg (Fasted): Phase I | Alectinib 460 mg (Fed): Phase I | Alectinib 600 mg (Fed): Phase I (20/40/150 mg) | Alectinib 760 mg (Fed): Phase I | Alectinib 900 mg (Fed): Phase I (20/40/150 mg) | Alectinib 600 mg (Fed): Phase II
Started | 7 | 7 | 13 | 7 | 13 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 7 | 13 | 7 | 13 | 0
Not completed — Death | 7 | 4 | 6 | 2 | 9 | 0
Not completed — Alive in Survival Follow-up | 0 | 2 | 4 | 5 | 4 | 0
Not completed — Lost to Follow-up | 0 | 1 | 3 | 0 | 0 | 0
Period: Phase II
Arm/Group | Alectinib 300 mg (Fasted): Phase I | Alectinib 460 mg (Fed): Phase I | Alectinib 600 mg (Fed): Phase I (20/40/150 mg) | Alectinib 760 mg (Fed): Phase I | Alectinib 900 mg (Fed): Phase I (20/40/150 mg) | Alectinib 600 mg (Fed): Phase II
Started | 0 | 0 | 0 | 0 | 0 | 87
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 87
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 45
Not completed — Alive in Survival Follow-up | 0 | 0 | 0 | 0 | 0 | 29
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 13

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any dose of alectinib.
Groups:
- Alectinib 300 mg (Fasted): Phase I: Participants received single dose of 20 or 40 mg alectinib capsules orally to make a dose of 240 or 300 mg on Cycle 1 Day -3 and then received 300 mg BID dose for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
- Alectinib 600 mg (Fed): Phase II: Participants received 600 mg alectinib capsules orally BID from Cycle 1 Day 1 for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
- Total: Total of all reporting groups
Arm/Group | Alectinib 300 mg (Fasted): Phase I | Alectinib 460 mg (Fed): Phase I | Alectinib 600 mg (Fed): Phase I (20/40/150 mg) | Alectinib 760 mg (Fed): Phase I | Alectinib 900 mg (Fed): Phase I (20/40/150 mg) | Alectinib 600 mg (Fed): Phase II | Total
Number analyzed (Participants) | 7 | 7 | 13 | 7 | 13 | 87 | 134
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 12 | 7 | 10 | 71 | 113
  >=65 years | 0 | 1 | 1 | 0 | 3 | 16 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 3 | 2 | 9 | 48 | 68
  Male | 5 | 3 | 10 | 5 | 4 | 39 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs): Phase I
Description: The DLTs were defined as any which included Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with bleeding or Grade 4 neutropenia continuing for greater than equal to (>=) 7 consecutive days, non-hematological toxicity of Grade 3 or higher (excluding transient electrolyte abnormalities, diarrhea, nausea, and vomiting that recovers to Grade 2 or lower with appropriate treatment and participants having Grade 2 aspartate transaminase (AST) and/or alanine transaminase (ALT) at baseline must have Grade 3 AST/ALT for 7 days or Grade 4 AST/ALT to be considered a DLT), and adverse events (AEs) that required suspension of treatment for a total of >=7 days which the Investigator could not rule out as been related to alectinib.
Time Frame: Throughout Cycle 1 of Phase I (21 days)
Population: Phase I safety population
Measure: Number; unit: participants
Arm/Group | Alectinib 300 mg (Fasted): Phase I | Alectinib 460 mg (Fed): Phase I | Alectinib 600 mg (Fed): Phase I (20/40/150 mg) | Alectinib 760 mg (Fed): Phase I | Alectinib 900 mg (Fed): Phase I (20/40/150 mg)
Number analyzed (Participants) | 7 | 7 | 13 | 7 | 13
participants | 0 | 0 | 0 | 0 | 2

2. Primary Outcome: Recommended Phase II Dose (RP2D): Phase I
Description: RP2D was defined as the highest dose with acceptable toxicity as determined from Phase I of the study.
Time Frame: Throughout Cycle 1 of Phase I (21 days)
Population: Phase I safety population
Measure: Number; unit: mg
Groups:
- Alectinib: Phase I: Participants received single dose of 20 or 40 or 150 mg alectinib capsules orally to make a dose of 240, 300, 460, 600, 760, or 900 mg on Cycle 1 Day -3 and then received 600 mg BID dose for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
Arm/Group | Alectinib: Phase I
Number analyzed (Participants) | 47
mg | 600

3. Primary Outcome: Percentage of Participants With Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) by Independent Review Committee (IRC): Phase II
Description: Percentage of participants with objective response as assessed by IRC was defined as the percentage of responders in the response evaluable population, where responders were defined as participants determined to have a best overall response of complete response (CR) or partial response (PR) based on the RECIST v1.1 criteria. CR: disappearance of all target and non-target lesions (TLs) and normalization of tumor markers. Pathological lymph nodes must have short axis measures less than (<) 10 millimeter (mm). PR: at least a 30 percent (%) decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of TLs, taking as reference the baseline sum of diameters. CR and PR were to be confirmed by repeat assessments >=4 weeks after initial documentation. Clopper-Pearson method was used to calculate 95% confidence interval (CI).
Time Frame: Cycle 1 Day 1 up to 194 weeks (assessed at every 6 weeks from Cycle 1 Day 1, at Cycles 2, 4, and 6 between Days 14-21, and every 3 cycles thereafter) (1 cycle = 21 days)
Population: Phase II Response evaluable (RE) population comprised all Phase II participants with measurable disease at baseline who had a baseline tumor assessment and received at least one dose of alectinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 67
percentage of participants | 52.2 [39.67 to 64.60]
Statistical Analysis 1: Comparison: Alectinib 600 mg (Fed): Phase II; Test type: Superiority; p = 0.0056, Exact Clopper-Pearson CI, 2 sided — Tests null hypothesis that the response rate is equal to 35% versus the alternative hypothesis that the response rate is not equal to 35%

4. Secondary Outcome: Percentage of Participants With Objective Response According to RECIST v1.1 by Investigator: Phase I
Description: Percentage of participants with objective response as assessed by Investigator was defined as the percentage of responders in the response evaluable population, where responders were defined as participants determined to have a best overall response of CR or PR based on the RECIST v1.1 criteria. CR: disappearance of all target and non-TLs and normalization of tumor markers. Pathological lymph nodes must have short axis measures <10 mm. PR: at least a 30% decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of TLs, taking as reference the baseline sum of diameters. CR and PR were to be confirmed by repeat assessments >=4 weeks after initial documentation. Clopper-Pearson method was used to calculate 95% CI. Data for this outcome were reported for 'alectinib 600 mg' and 'alectinib other than 600 mg' groups as planned.
Time Frame: Every 6 weeks from Cycle 1 Day 1, at Cycles 2, 4, and 6 between Days 14-21, and every 3 cycles thereafter (assessed up to 194 weeks) (1 cycle = 21 days)
Population: Phase I RE population comprised all Phase I participants with measurable disease at baseline who had a baseline tumor assessment and received at least one dose of alectinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Alectinib Other Than 600 mg (Fasted/Fed): Phase I: Participants received single dose of 20 or 40 or 150 mg alectinib capsules orally to make a dose of 240, 300, 460, 760, or 900 mg on Cycle 1 Day -3 and then received 300, 460, 760, or 900 mg BID dose for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
Arm/Group | Alectinib 600 mg (Fed): Phase I (20/40/150 mg) | Alectinib Other Than 600 mg (Fasted/Fed): Phase I
Number analyzed (Participants) | 13 | 34
percentage of participants | 69.2 [38.57 to 90.91] | 55.9 [37.89 to 72.81]
Statistical Analysis 1: Comparison: Alectinib 600 mg (Fed): Phase I (20/40/150 mg); Test type: Superiority; p = 0.0251, Exact Clopper-Pearson CI, 2 sided — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Alectinib Other Than 600 mg (Fasted/Fed): Phase I; Test type: Superiority; p = 0.0203, Exact Clopper-Pearson CI, 2 sided — [p-value comment as in outcome 3, analysis 1]

5. Secondary Outcome: Duration of Response (DOR) According to RECIST v1.1 by Investigator: Phase I
Description: DOR was defined for responders (CR or PR) as the time from when response was first documented, to first documented disease progression (according to RECIST v1.1) or death (whichever occurred first). Participants who did not progress or did not die after they had a response were censored at date of their last tumor measurement. Progressive disease (PD): at least 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions. Refer "Outcome Measure 2" for the definition of CR and PR. The median time to the event was estimated using the methodology of Kaplan-Meier. Brookmeyer-Crowley method was used to calculate 95% CI. Data for this outcome were reported for 'alectinib 600 mg' and 'alectinib other than 600 mg' groups as planned.
Time Frame: as for outcome 4
Population: Phase I RE population. 'Overall Number of Participants Analyzed' = participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib 600 mg (Fed): Phase I (20/40/150 mg) | Alectinib Other Than 600 mg (Fasted/Fed): Phase I
Number analyzed (Participants) | 9 | 19
months | 12.2 [4.9 to 20.9] | 11.0 [6.3 to 14.8]

6. Secondary Outcome: Percentage of Participants With Objective Response According to RECIST v1.1 by Investigator: Phase II
Description: Percentage of participants with objective response as assessed by Investigator was defined as the percentage of responders in the response evaluable population, where responders were defined as participants determined to have a best overall response of CR or PR based on the RECIST v1.1 criteria. CR: disappearance of all target and non-TLs and normalization of tumor markers. Pathological lymph nodes must have short axis measures <10 mm. PR: at least a 30% decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of TLs, taking as reference the baseline sum of diameters. CR and PR were to be confirmed by repeat assessments >=4 weeks after initial documentation. Clopper-Pearson method was used to calculate 95% CI.
Time Frame: as for outcome 4
Population: Phase II RE population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 87
percentage of participants | 52.9 [41.87 to 63.67]
Statistical Analysis 1: Comparison: Alectinib 600 mg (Fed): Phase II; Test type: Superiority; p = 0.0010, Exact Clopper-Pearson CI, 2 sided — [p-value comment as in outcome 3, analysis 1]

7. Secondary Outcome: Percentage of Participants With Disease Control According to RECIST v1.1 by Investigator: Phase II
Description: Disease control rate assessed according to RECIST v1.1 was defined as the percentage of participants with a best overall response of CR, PR, or stable disease (SD) lasting for at least 12 weeks, after the first dose of alectinib. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum of diameters on study. PD: at least 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions. CR: disappearance of all target and non-TLs and normalization of tumor markers. Pathological lymph nodes must have short axis measures <10 mm. PR: at least a 30% decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of TLs, taking as reference the baseline sum of diameters. 95% CI for rate was constructed using Clopper-Pearson method.
Time Frame: as for outcome 4
Population: Phase II RE population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 87
percentage of participants | 66.7 [55.75 to 76.42]

8. Secondary Outcome: Percentage of Participants With Disease Progression According to RECIST v1.1 by IRC or Death : Phase II
Description: Percentage of participants with disease progression according to RECIST v1.1 by IRC is defined as the participants with at least 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions.
Time Frame: as for outcome 4
Population: Phase II safety population
Measure: Number; unit: percentage of participants
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 87
percentage of participants | 66.7

9. Secondary Outcome: Progression-Free Survival (PFS) According to RECIST v1.1 by IRC: Phase II
Description: PFS was defined as the time between first dose of alectinib and date of first documented disease progression according to RECIST v1.1 or death, whichever occurred first. Participants who have neither progressed nor died at the time of the last clinical cut-off or who lost to follow-up were censored at the date of the last tumor assessment showing no progression of disease either during the study treatment or during follow-up. Participants with no post-baseline assessments were censored at the date of first dose. Progression of disease is defined as at least 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions. The median time to the event was estimated using the methodology of Kaplan-Meier. Brookmeyer-Crowley method was used to calculate 95% CI.
Time Frame: as for outcome 4
Population: Phase II safety population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 87
months | 8.2 [6.3 to 12.6]

10. Secondary Outcome: Percentage of Participants With Disease Progression According to RECIST v1.1 by Investigator or Death : Phase II
Description: Percentage of participants with disease progression according to RECIST v1.1 by investigator is defined as the participants with at least 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions.
Time Frame: as for outcome 4
Population: Phase II safety population
Measure: Number; unit: percentage of participants
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 87
percentage of participants | 70.1

11. Secondary Outcome: PFS According to RECIST v1.1 by Investigator: Phase II
Description: as for outcome 9
Time Frame: as for outcome 4
Population: Phase II RE population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 87
months | 8.4 [5.5 to 12.7]

12. Secondary Outcome: Percentage of Participants Who Died Due to Any Cause: Phase II
Time Frame: Baseline up to death (any cause) (maximum follow up 284 weeks)
Population: Phase II safety population
Measure: Number; unit: percentage of participants
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 87
percentage of participants | 51.7

13. Secondary Outcome: Overall Survival (OS) Time: Phase II
Description: OS was defined as the time between date of first dose and date of death due to any cause. Participants without an event were censored at the date last known to be alive. Participants without any follow-up information were censored at the date of first dose. The median time to the event was estimated using the methodology of Kaplan-Meier. Brookmeyer-Crowley method was used to calculate 95% CI.
Time Frame: Baseline up to death (any cause) (maximum follow up 284 weeks)
Population: Phase II safety population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 87
months | 27.9 [17.2 to NA] — Upper limit of 95% CI was not estimable due to low number of events and longer observation time.

14. Secondary Outcome: DOR According to RECIST v1.1 by IRC: Phase II
Description: DOR was defined for responders (CR or PR) as the time from when response was first documented, to first documented disease progression (according to RECIST v1.1) or death (whichever occurred first). Participants who did not progress or did not die after they had a response were censored at date of their last tumor measurement. Progressive disease (PD): at least 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions. Refer "Outcome Measure 2" for the definition of CR and PR. The median time to the event was estimated using the methodology of Kaplan-Meier. Brookmeyer-Crowley method was used to calculate 95% CI.
Time Frame: as for outcome 4
Population: Phase II RE population. 'Overall Number of Participants Analyzed' = participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 35
months | 14.9 [6.9 to NA] — Upper limit of 95% CI was not estimable due to low number of events and longer observation time.

15. Secondary Outcome: DOR According to RECIST v1.1 by Investigator: Phase II
Description: as for outcome 14
Time Frame: as for outcome 4
Population: Phase II RE population. 'Overall Number of Participants Analyzed' = participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 46
months | 13.3 [8.8 to 18.2]

16. Secondary Outcome: Percentage of Participants With Central Nervous System Objective Response (COR) According to RECIST v1.1 by IRC: Phase II
Description: COR rate (CORR) was defined as the percentage of participants who had a CR or PR of the baseline central nervous system (CNS) lesions, based on RECIST v.1.1. CNS responses according to RECIST v1.1 did not have to be confirmed. CR was defined as disappearance of all CNS lesions. PR was defined as >=30% decrease in the sum of diameters of measurable CNS lesions (taking as reference the baseline sum of diameters). 95% CI was computed using the Clopper-Pearson method.
Time Frame: as for outcome 4
Population: Phase II safety population. 'Overall Number of Participants Analyzed' = participants with measurable CNS lesions at baseline based on RECIST v1.1 according to IRC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 16
percentage of participants | 75.0 [47.62 to 92.73]

17. Secondary Outcome: Percentage of Participants With COR According to Response Assessment in Neuro-Oncology (RANO) Criteria by IRC: Phase II
Description: CORR was defined as the percentage of participants who had a CR or PR according to RANO criteria of the baseline CNS lesions. As per RANO criteria, CR was defined as disappearance of all enhancing measurable and non-measurable disease, and no new lesions along with stable or clinically improved status, participants off corticosteroids (or on physiologic replacement doses only) and stable or improved non enhancing T2/FLAIR lesions; PR was defined as 50% or more decrease in sum of the products of the diameters (SPD) of measurable enhancing measurable lesions, no new lesion along with stable or clinically improved status, participants off corticosteroids (or on physiologic replacement doses only) and no progression of non-measurable disease (enhancing and non-enhancing T2/FLAIR lesions. Clopper-Pearson method was used to calculate 95% CI.
Time Frame: as for outcome 4
Population: Phase II safety population. 'Overall Number of Participants Analyzed' = participants with measurable CNS lesions at baseline according to RANO criteria by IRC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 11
percentage of participants | 54.5 [23.38 to 83.25]

18. Secondary Outcome: CNS Duration of Response (CDOR) According to RECIST v1.1 by IRC: Phase II
Description: CDOR was defined for CNS responders as the time from the first observation of a CNS response of CR or PR until first observation of CNS progression or death from any cause. An analysis by IRC using RECIST v1.1 was performed. PD: at least 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and absolute increase of at least 5 mm, or presence of new lesions. CR was defined as disappearance of all CNS lesions. PR was defined as >=30% decrease in the sum of diameters of measurable CNS lesions (taking as reference the baseline sum of diameters). The median time to the event was estimated using the methodology of Kaplan-Meier. Brookmeyer-Crowley method was used to calculate 95% CI.
Time Frame: as for outcome 4
Population: Phase II safety population. 'Overall Number of Participants Analyzed' = participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 12
months | 11.1 [5.8 to NA] — Upper limit of 95% CI was not estimable due to low number of events and longer observation time.

19. Secondary Outcome: CDOR According to RANO Criteria by IRC: Phase II
Description: CDOR was defined as the time from the first observation of a CNS response of CR or PR according to RANO criteria until first observation of CNS progression or death from any cause. An analysis by RANO criteria was performed. Definitions of CR or PR as per RANO was included in description of Outcome Measure 17. As per RANO criteria, progression was defined as 25% or more increase in SPD of measurable enhancing (measurable) compared to the best response after initiation of therapy or Screening; increase (significant) in non-enhancing T2/FLAIR lesions, not attributable to other non-tumor causes; any new lesions; and clinical deterioration (not attributable to other non-tumor causes and not due to steroid decrease) and clear worsening of neurological status with respect to the previous timepoint. The median time to the event was estimated using the methodology of Kaplan-Meier. Brookmeyer-Crowley method was used to calculate 95% CI.
Time Frame: as for outcome 4
Population: Phase II safety population. 'Overall Number of Participants Analyzed' = participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 6
months | 12.1 [11.1 to NA] — Upper limit of 95% CI was not estimable due to low number of events and longer observation time.

20. Secondary Outcome: Percentage of Participants With CNS Progression According to RECIST v1.1 by IRC: Phase II
Description: CNS disease progression was defined as a new CNS lesion or progression of pre-existing CNS lesions according to RECIST v1.1. PD: at least 20% increase in the sum of diameters of target lesions compared to the smallest sum of diameters on-study and absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions.
Time Frame: as for outcome 4
Population: Phase II safety population. 'Overall Number of Participants Analyzed' = participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 16
percentage of participants | 0 [0.00 to 20.59]

21. Secondary Outcome: Percentage of Participants With CNS Progression According to RANO Criteria by IRC: Phase II
Description: CNS disease progression was defined as a new CNS lesion or progression of pre-existing CNS lesions according to RANO criteria. As per RANO criteria, progression was defined as 25% or more increase in SPD of measurable enhancing (measurable) compared to the best response after initiation of therapy or Screening; increase (significant) in non-enhancing T2/FLAIR lesions, not attributable to other non-tumor causes; any new lesions; and clinical deterioration (not attributable to other non-tumor causes and not due to steroid decrease).
Time Frame: as for outcome 4
Population: Data were not estimable due to low number of responders and longer observation time.
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 0

22. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) After Single Dose of Alectinib: Phase I
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 4, 6, 8, 10, 24, 32 and 48 hours post-dose on Cycle 1 Day -3 (1 cycle = 21 days)
Population: Phase I pharmacokinetic (PK) evaluable population included all participants who received any dose of alectinib and who had at least one post-baseline PK sample available. 'Overall Number of Participants Analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- Alectinib 240 mg Once and 300 mg BID (Fasted): Phase I: Participants (in fasting condition) received single dose of 20 or 40 mg alectinib capsules orally to make a dose of 240 mg on Cycle 1 Day -3 and then received 300 mg BID dose for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
- Alectinib 240 mg Once and 300 mg BID (Fed): Phase I: Participants (in non-fasting condition) received single dose of 20 or 40 mg alectinib capsules orally to make a dose of 240 mg on Cycle 1 Day -3 and then received 300 mg BID dose for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
- Alectinib 300 mg (Fasted): Phase I: Participants received single dose of 20 or 40 mg alectinib capsules orally to make a dose of 300 mg on Cycle 1 Day -3 and then received 300 mg BID dose for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
- Alectinib 600 mg (Fed): Phase I (20/40 mg): Participants received single dose of 20 or 40 mg alectinib capsules orally to make a dose of 600 mg on Cycle 1 Day -3 and then received 600 mg BID dose for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
- Alectinib 600 mg (Fed): Phase I (150 mg): Participants received single dose of 150 mg alectinib capsules orally to make a dose of 600 mg on Cycle 1 Day -3 and then received 600 mg BID dose for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
- Alectinib 900 mg (Fed): Phase I (20/40 mg): Participants received single dose of 20 or 40 mg alectinib capsules orally to make a dose of 900 mg on Cycle 1 Day -3 and then received 900 mg BID dose for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
- Alectinib 900 mg (Fed): Phase I (150 mg): Participants received single dose of 150 mg alectinib capsules orally to make a dose of 900 mg on Cycle 1 Day -3 and then received 900 mg BID for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
Arm/Group | Alectinib 240 mg Once and 300 mg BID (Fasted): Phase I | Alectinib 240 mg Once and 300 mg BID (Fed): Phase I | Alectinib 300 mg (Fasted): Phase I | Alectinib 460 mg (Fed): Phase I | Alectinib 600 mg (Fed): Phase I (20/40 mg) | Alectinib 600 mg (Fed): Phase I (150 mg) | Alectinib 760 mg (Fed): Phase I | Alectinib 900 mg (Fed): Phase I (20/40 mg) | Alectinib 900 mg (Fed): Phase I (150 mg)
Number analyzed (Participants) | 3 | 1 | 3 | 7 | 6 | 6 | 7 | 7 | 6
nanograms per milliliter (ng/mL) | 73.5 (12.4) | 87.7 | 45.3 (9.24) | 142.00 (71.4) | 158.0 (67.2) | 186.0 (43.1) | 257.0 (83.1) | 186.0 (120.0) | 295.0 (131.0)

23. Secondary Outcome: Cmax After Multiple Dose of Alectinib: Phase I
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 4, 6, 8 and 10 hours post-dose on Cycle 2 Day 1 (1 cycle = 21 days)
Population: Phase I PK evaluable population. 'Overall Number of Participants Analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alectinib 300 mg (Fasted): Phase I | Alectinib 460 mg (Fed): Phase I | Alectinib 600 mg (Fed): Phase I (20/40 mg) | Alectinib 600 mg (Fed): Phase I (150 mg) | Alectinib 760 mg (Fed): Phase I | Alectinib 900 mg (Fed): Phase I (20/40 mg) | Alectinib 900 mg (Fed): Phase I (150 mg)
Number analyzed (Participants) | 6 | 7 | 5 | 6 | 5 | 7 | 4
ng/mL | 259 (79.0) | 618 (165) | 765 (176) | 670 (360) | 733 (98.0) | 1140 (448) | 1200 (311)

24. Secondary Outcome: Area Under the Plasma Concentration (AUC) Versus Time Curve Extrapolated to Infinity (AUCinf) After Single Dose of Alectinib: Phase I
Description: AUCinf = AUC from time zero (pre-dose) to extrapolated infinite time. It is obtained from AUC (0- t) plus AUC (t-inf).
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 4, 6, 8, 10, 24, 32 and 48 hours post-dose on Cycle 1 Day -3 (1 cycle = 21 days)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Alectinib 240 mg Once and 300 mg BID (Fasted): Phase I | Alectinib 240 mg Once and 300 mg BID (Fed): Phase I | Alectinib 300 mg (Fasted): Phase I | Alectinib 460 mg (Fed): Phase I | Alectinib 600 mg (Fed): Phase I (20/40 mg) | Alectinib 600 mg (Fed): Phase I (150 mg) | Alectinib 760 mg (Fed): Phase I | Alectinib 900 mg (Fed): Phase I (20/40 mg) | Alectinib 900 mg (Fed): Phase I (150 mg)
Number analyzed (Participants) | 3 | 1 | 3 | 7 | 6 | 6 | 7 | 7 | 6
hour*ng/mL | 1360 (436) | 858 | 1030 (481) | 3280 (2240) | 3310 (1110) | 3190 (1510) | 4090 (1680) | 3730 (2310) | 7790 (6210)

25. Secondary Outcome: AUC From Time Zero to Last Measurable Concentration (AUClast) After Multiple Dose of Alectinib: Phase I
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 4, 6, 8 and 10 hours post-dose on Cycle 2 Day 1 (1 cycle = 21 days)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Alectinib 300 mg (Fasted): Phase I | Alectinib 460 mg (Fed): Phase I | Alectinib 600 mg (Fed): Phase I (20/40 mg) | Alectinib 600 mg (Fed): Phase I (150 mg) | Alectinib 760 mg (Fed): Phase I | Alectinib 900 mg (Fed): Phase I (20/40 mg) | Alectinib 900 mg (Fed): Phase I (150 mg)
Number analyzed (Participants) | 6 | 7 | 5 | 6 | 5 | 7 | 4
hour*ng/mL | 1800 (562) | 4510 (1700) | 5970 (1140) | 5300 (3180) | 5780 (1020) | 9800 (4660) | 9500 (2670)

26. Secondary Outcome: Ctrough After Multiple Dose of Alectinib: Phase II
Time Frame: Pre-dose (0 hour) on Day 1 of Cycles 2, Cycle 3, Cycle 4, Cycle 5 (1 cycle = 21 days)
Population: Phase II PK evaluable population. 'Overall Number of Participants Analyzed' = participants evaluable for this outcome measure. 'Number Analyzed' = number of participants evaluable at the specified timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 61
ng/mL
  Cycle 2 Day 1 | 473 (277)
  Cycle 3 Day 1: number analyzed (Participants) | 51
  Cycle 3 Day 1 | 521 (272)
  Cycle 4 Day 1: number analyzed (Participants) | 52
  Cycle 4 Day 1 | 538 (279)
  Cycle 5 Day 1: number analyzed (Participants) | 45
  Cycle 5 Day 1 | 538 (226)

27. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30): Phase II
Description: EORTC QLQ-C30 included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions used 4-point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale [1 'very poor' to 7 'Excellent']). Scores were averaged and transformed to lie between 0-100 scale; for each of the symptom scales, higher score=better level of functioning, lower score indicates lower level of functioning. 'Baseline' category for any parameter below (e.g. Global health status/QoL [quality of life]) represents absolute data at baseline. QoL=quality of life
Time Frame: Baseline, Weeks 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69, 72, 75, 78, 81, 84, 87, 90, 93, 96, 99, 105, 111, 117, last visit (up to 194 weeks)
Population: Phase II safety population. 'Overall Number of Participants Analyzed' = participants evaluable for this outcome measure. 'Number Analyzed' = number of participants evaluable at the specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 79
units on a scale
  Global health status/QoL: Baseline | 53.59 (24.27)
  Global health status/QoL: Week 6: number analyzed (Participants) | 64
  Global health status/QoL: Week 6 | 15.89 (25.66)
  Global health status/QoL: Week 9: number analyzed (Participants) | 1
  Global health status/QoL: Week 9 | 0.00
  Global health status/QoL: Week 12: number analyzed (Participants) | 54
  Global health status/QoL: Week 12 | 18.83 (23.41)
  Global health status/QoL: Week 15: number analyzed (Participants) | 1
  Global health status/QoL: Week 15 | 0.00
  Global health status/QoL: Week 18: number analyzed (Participants) | 49
  Global health status/QoL: Week 18 | 15.65 (23.73)
  Global health status/QoL: Week 21: number analyzed (Participants) | 1
  Global health status/QoL: Week 21 | 0.00
  Global health status/QoL: Week 24: number analyzed (Participants) | 41
  Global health status/QoL: Week 24 | 15.65 (20.77)
  Global health status/QoL: Week 27: number analyzed (Participants) | 2
  Global health status/QoL: Week 27 | 0.00 (0.00)
  Global health status/QoL: Week 30: number analyzed (Participants) | 39
  Global health status/QoL: Week 30 | 13.03 (19.57)
  Global health status/QoL: Week 33: number analyzed (Participants) | 3
  Global health status/QoL: Week 33 | -5.56 (9.62)
  Global health status/QoL: Week 36: number analyzed (Participants) | 38
  Global health status/QoL: Week 36 | 12.28 (20.57)
  Global health status/QoL: Week 39: number analyzed (Participants) | 2
  Global health status/QoL: Week 39 | 4.17 (5.89)
  Global health status/QoL: Week 42: number analyzed (Participants) | 36
  Global health status/QoL: Week 42 | 10.19 (19.33)
  Global health status/QoL: Week 45: number analyzed (Participants) | 4
  Global health status/QoL: Week 45 | -10.42 (12.50)
  Global health status/QoL: Week 48: number analyzed (Participants) | 33
  Global health status/QoL: Week 48 | 11.11 (19.06)
  Global health status/QoL: Week 51: number analyzed (Participants) | 2
  Global health status/QoL: Week 51 | 12.50 (17.68)
  Global health status/QoL: Week 54: number analyzed (Participants) | 31
  Global health status/QoL: Week 54 | 9.95 (16.86)
  Global health status/QoL: Week 57: number analyzed (Participants) | 5
  Global health status/QoL: Week 57 | -3.33 (21.73)
  Global health status/QoL: Week 60: number analyzed (Participants) | 30
  Global health status/QoL: Week 60 | 10.28 (19.54)
  Global health status/QoL: Week 63: number analyzed (Participants) | 3
  Global health status/QoL: Week 63 | 11.11 (19.25)
  Global health status/QoL: Week 66: number analyzed (Participants) | 26
  Global health status/QoL: Week 66 | 15.06 (17.80)
  Global health status/QoL: Week 69: number analyzed (Participants) | 4
  Global health status/QoL: Week 69 | 12.50 (15.96)
  Global health status/QoL: Week 72: number analyzed (Participants) | 23
  Global health status/QoL: Week 72 | 8.33 (18.12)
  Global health status/QoL: Week 75: number analyzed (Participants) | 2
  Global health status/QoL: Week 75 | 16.67 (23.57)
  Global health status/QoL: Week 78: number analyzed (Participants) | 21
  Global health status/QoL: Week 78 | 10.32 (16.44)
  Global health status/QoL: Week 81: number analyzed (Participants) | 2
  Global health status/QoL: Week 81 | 16.67 (23.57)
  Global health status/QoL: Week 84: number analyzed (Participants) | 13
  Global health status/QoL: Week 84 | 10.90 (14.98)
  Global health status/QoL: Week 87: number analyzed (Participants) | 3
  Global health status/QoL: Week 87 | 11.11 (19.25)
  Global health status/QoL: Week 90: number analyzed (Participants) | 8
  Global health status/QoL: Week 90 | 4.17 (11.79)
  Global health status/QoL: Week 93: number analyzed (Participants) | 2
  Global health status/QoL: Week 93 | -29.17 (41.25)
  Global health status/QoL: Week 96: number analyzed (Participants) | 3
  Global health status/QoL: Week 96 | 0.00 (22.05)
  Global health status/QoL: Week 99: number analyzed (Participants) | 1
  Global health status/QoL: Week 99 | -16.67
  Global health status/QoL: Week 105: number analyzed (Participants) | 1
  Global health status/QoL: Week 105 | -16.67
  Global health status/QoL: Week 111: number analyzed (Participants) | 1
  Global health status/QoL: Week 111 | 0.00
  Global health status/QoL: Week 117: number analyzed (Participants) | 1
  Global health status/QoL: Week 117 | 0.00
  Global health status/QoL: Last visit: number analyzed (Participants) | 73
  Global health status/QoL: Last visit | 7.99 (21.27)
  Physical functioning: Baseline | 69.96 (24.43)
  Physical functioning: Week 6: number analyzed (Participants) | 64
  Physical functioning: Week 6 | 4.69 (17.44)
  Physical functioning: Week 9: number analyzed (Participants) | 1
  Physical functioning: Week 9 | 0.00
  Physical functioning: Week 12: number analyzed (Participants) | 54
  Physical functioning: Week 12 | 4.20 (22.37)
  Physical functioning: Week 15: number analyzed (Participants) | 1
  Physical functioning: Week 15 | 0.00
  Physical functioning: Week 18: number analyzed (Participants) | 51
  Physical functioning: Week 18 | 7.58 (18.23)
  Physical functioning: Week 21: number analyzed (Participants) | 1
  Physical functioning: Week 21 | 0.00
  Physical functioning: Week 24: number analyzed (Participants) | 42
  Physical functioning: Week 24 | 4.13 (16.33)
  Physical functioning: Week 27: number analyzed (Participants) | 2
  Physical functioning: Week 27 | 3.33 (4.71)
  Physical functioning: Week 30: number analyzed (Participants) | 39
  Physical functioning: Week 30 | 2.22 (17.39)
  Physical functioning: Week 33: number analyzed (Participants) | 3
  Physical functioning: Week 33 | 0.00 (13.33)
  Physical functioning: Week 36: number analyzed (Participants) | 38
  Physical functioning: Week 36 | 4.21 (18.10)
  Physical functioning: Week 39: number analyzed (Participants) | 2
  Physical functioning: Week 39 | 3.33 (14.14)
  Physical functioning: Week 42: number analyzed (Participants) | 36
  Physical functioning: Week 42 | 6.85 (18.89)
  Physical functioning: Week 45: number analyzed (Participants) | 4
  Physical functioning: Week 45 | -3.33 (22.11)
  Physical functioning: Week 48: number analyzed (Participants) | 33
  Physical functioning: Week 48 | 5.25 (16.81)
  Physical functioning: Week 51: number analyzed (Participants) | 2
  Physical functioning: Week 51 | 0.00 (18.86)
  Physical functioning: Week 54: number analyzed (Participants) | 32
  Physical functioning: Week 54 | 6.67 (18.32)
  Physical functioning: Week 57: number analyzed (Participants) | 5
  Physical functioning: Week 57 | 0.00 (20.55)
  Physical functioning: Week 60: number analyzed (Participants) | 30
  Physical functioning: Week 60 | 7.56 (22.67)
  Physical functioning: Week 63: number analyzed (Participants) | 3
  Physical functioning: Week 63 | -6.67 (11.55)
  Physical functioning: Week 66: number analyzed (Participants) | 26
  Physical functioning: Week 66 | 8.97 (19.13)
  Physical functioning: Week 69: number analyzed (Participants) | 4
  Physical functioning: Week 69 | 8.33 (16.67)
  Physical functioning: Week 72: number analyzed (Participants) | 23
  Physical functioning: Week 72 | 4.20 (22.70)
  Physical functioning: Week 75: number analyzed (Participants) | 2
  Physical functioning: Week 75 | 0.00 (0.00)
  Physical functioning: Week 78: number analyzed (Participants) | 21
  Physical functioning: Week 78 | 6.98 (19.83)
  Physical functioning: Week 81: number analyzed (Participants) | 2
  Physical functioning: Week 81 | 0.00 (0.00)
  Physical functioning: Week 84: number analyzed (Participants) | 13
  Physical functioning: Week 84 | 3.08 (21.71)
  Physical functioning: Week 87: number analyzed (Participants) | 3
  Physical functioning: Week 87 | -6.67 (11.55)
  Physical functioning: Week 90: number analyzed (Participants) | 8
  Physical functioning: Week 90 | 7.50 (18.32)
  Physical functioning: Week 93: number analyzed (Participants) | 2
  Physical functioning: Week 93 | -26.67 (28.28)
  Physical functioning: Week 96: number analyzed (Participants) | 3
  Physical functioning: Week 96 | 33.33 (11.55)
  Physical functioning: Week 99: number analyzed (Participants) | 1
  Physical functioning: Week 99 | -6.67
  Physical functioning: Week 105: number analyzed (Participants) | 1
  Physical functioning: Week 105 | 0.00
  Physical functioning: Week 111: number analyzed (Participants) | 1
  Physical functioning: Week 111 | 0.00
  Physical functioning: Week 117: number analyzed (Participants) | 1
  Physical functioning: Week 117 | 0.00
  Physical functioning: Last visit: number analyzed (Participants) | 73
  Physical functioning: Last visit | 2.28 (21.64)
  Role functioning: Baseline | 58.86 (34.06)
  Role functioning: Week 6: number analyzed (Participants) | 64
  Role functioning: Week 6 | 14.84 (32.00)
  Role functioning: Week 9: number analyzed (Participants) | 1
  Role functioning: Week 9 | 0.00
  Role functioning: Week 12: number analyzed (Participants) | 54
  Role functioning: Week 12 | 12.65 (32.69)
  Role functioning: Week 15: number analyzed (Participants) | 1
  Role functioning: Week 15 | 0.00
  Role functioning: Week 18: number analyzed (Participants) | 51
  Role functioning: Week 18 | 12.42 (31.94)
  Role functioning: Week 21: number analyzed (Participants) | 1
  Role functioning: Week 21 | 0.00
  Role functioning: Week 24: number analyzed (Participants) | 42
  Role functioning: Week 24 | 8.73 (27.85)
  Role functioning: Week 27: number analyzed (Participants) | 2
  Role functioning: Week 27 | -8.33 (11.79)
  Role functioning: Week 30: number analyzed (Participants) | 39
  Role functioning: Week 30 | 9.83 (24.70)
  Role functioning: Week 33: number analyzed (Participants) | 3
  Role functioning: Week 33 | -33.33 (33.33)
  Role functioning: Week 36: number analyzed (Participants) | 38
  Role functioning: Week 36 | 9.65 (24.70)
  Role functioning: Week 39: number analyzed (Participants) | 2
  Role functioning: Week 39 | -33.33 (0.00)
  Role functioning: Week 42: number analyzed (Participants) | 36
  Role functioning: Week 42 | 6.48 (28.81)
  Role functioning Week 45: number analyzed (Participants) | 4
  Role functioning Week 45 | -20.83 (15.96)
  Role functioning: Week 48: number analyzed (Participants) | 32
  Role functioning: Week 48 | 10.94 (24.54)
  Role functioning: Week 51: number analyzed (Participants) | 2
  Role functioning: Week 51 | -16.67 (23.57)
  Role functioning: Week 54: number analyzed (Participants) | 32
  Role functioning: Week 54 | 7.29 (24.30)
  Role functioning: Week 57: number analyzed (Participants) | 5
  Role functioning: Week 57 | -13.33 (18.26)
  Role functioning: Week 60: number analyzed (Participants) | 30
  Role functioning: Week 60 | 8.89 (27.24)
  Role functioning: Week 63: number analyzed (Participants) | 3
  Role functioning: Week 63 | -5.56 (9.62)
  Role functioning: Week 66: number analyzed (Participants) | 26
  Role functioning: Week 66 | 8.97 (29.90)
  Role functioning: Week 69: number analyzed (Participants) | 4
  Role functioning: Week 69 | -16.67 (33.33)
  Role functioning: Week 72: number analyzed (Participants) | 23
  Role functioning: Week 72 | 7.97 (27.46)
  Role functioning: Week 75: number analyzed (Participants) | 2
  Role functioning: Week 75 | 0.00 (0.00)
  Role functioning: Week 78: number analyzed (Participants) | 21
  Role functioning: Week 78 | 9.52 (28.66)
  Role functioning: Week 81: number analyzed (Participants) | 2
  Role functioning: Week 81 | 0.00 (0.00)
  Role functioning: Week 84: number analyzed (Participants) | 13
  Role functioning: Week 84 | 5.13 (31.46)
  Role functioning: Week 87: number analyzed (Participants) | 3
  Role functioning: Week 87 | -11.11 (19.25)
  Role functioning: Week 90: number analyzed (Participants) | 8
  Role functioning: Week 90 | -4.17 (19.42)
  Role functioning: Week 93: number analyzed (Participants) | 2
  Role functioning: Week 93 | -41.67 (35.36)
  Role functioning: Week 96: number analyzed (Participants) | 3
  Role functioning: Week 96 | 11.11 (19.25)
  Role functioning: Week 99: number analyzed (Participants) | 1
  Role functioning: Week 99 | -16.67
  Role functioning: Week 105: number analyzed (Participants) | 1
  Role functioning: Week 105 | 0.00
  Role functioning: Week 111: number analyzed (Participants) | 1
  Role functioning: Week 111 | 0.00
  Role functioning: Week 117: number analyzed (Participants) | 1
  Role functioning: Week 117 | 0.00
  Role functioning: Last visit: number analyzed (Participants) | 73
  Role functioning: Last visit | 9.36 (34.47)
  Emotional functioning: Baseline | 73.49 (21.40)
  Emotional functioning: Week 6: number analyzed (Participants) | 64
  Emotional functioning: Week 6 | 7.99 (18.75)
  Emotional functioning: Week 9: number analyzed (Participants) | 1
  Emotional functioning: Week 9 | 0.00
  Emotional functioning: Week 12: number analyzed (Participants) | 54
  Emotional functioning: Week 12 | 11.01 (17.04)
  Emotional functioning: Week 15: number analyzed (Participants) | 1
  Emotional functioning: Week 15 | 0.00
  Emotional functioning: Week 18: number analyzed (Participants) | 49
  Emotional functioning: Week 18 | 13.44 (21.17)
  Emotional functioning: Week 21: number analyzed (Participants) | 1
  Emotional functioning: Week 21 | 0.00
  Emotional functioning: Week 24: number analyzed (Participants) | 41
  Emotional functioning: Week 24 | 10.37 (16.75)
  Emotional functioning: Week 27: number analyzed (Participants) | 2
  Emotional functioning: Week 27 | -4.17 (5.89)
  Emotional functioning: Week 30: number analyzed (Participants) | 39
  Emotional functioning: Week 30 | 9.40 (20.34)
  Emotional functioning: Week 33: number analyzed (Participants) | 3
  Emotional functioning: Week 33 | -30.56 (26.79)
  Emotional functioning: Week 36: number analyzed (Participants) | 38
  Emotional functioning: Week 36 | 7.89 (19.85)
  Emotional functioning: Week 39: number analyzed (Participants) | 2
  Emotional functioning: Week 39 | -4.17 (5.89)
  Emotional functioning: Week 42: number analyzed (Participants) | 36
  Emotional functioning: Week 42 | 7.41 (18.12)
  Emotional functioning Week 45: number analyzed (Participants) | 4
  Emotional functioning Week 45 | -6.25 (7.98)
  Emotional functioning: Week 48: number analyzed (Participants) | 33
  Emotional functioning: Week 48 | 6.73 (15.23)
  Emotional functioning: Week 51: number analyzed (Participants) | 2
  Emotional functioning: Week 51 | 0.00 (0.00)
  Emotional functioning: Week 54: number analyzed (Participants) | 31
  Emotional functioning: Week 54 | 3.49 (13.40)
  Emotional functioning: Week 57: number analyzed (Participants) | 5
  Emotional functioning: Week 57 | -6.67 (18.07)
  Emotional functioning: Week 60: number analyzed (Participants) | 30
  Emotional functioning: Week 60 | 3.33 (14.12)
  Emotional functioning: Week 63: number analyzed (Participants) | 3
  Emotional functioning: Week 63 | -11.11 (34.69)
  Emotional functioning: Week 66: number analyzed (Participants) | 26
  Emotional functioning: Week 66 | 5.45 (14.52)
  Emotional functioning: Week 69: number analyzed (Participants) | 4
  Emotional functioning: Week 69 | -8.33 (26.35)
  Emotional functioning: Week 72: number analyzed (Participants) | 23
  Emotional functioning: Week 72 | 5.07 (21.43)
  Emotional functioning: Week 75: number analyzed (Participants) | 2
  Emotional functioning: Week 75 | 8.33 (11.79)
  Emotional functioning: Week 78: number analyzed (Participants) | 21
  Emotional functioning: Week 78 | -1.19 (19.77)
  Emotional functioning: Week 81: number analyzed (Participants) | 2
  Emotional functioning: Week 81 | 4.17 (5.89)
  Emotional functioning: Week 84: number analyzed (Participants) | 13
  Emotional functioning: Week 84 | 1.28 (19.79)
  Emotional functioning: Week 87: number analyzed (Participants) | 3
  Emotional functioning: Week 87 | -11.11 (34.69)
  Emotional functioning: Week 90: number analyzed (Participants) | 8
  Emotional functioning: Week 90 | 1.04 (8.26)
  Emotional functioning: Week 93: number analyzed (Participants) | 2
  Emotional functioning: Week 93 | -12.50 (17.68)
  Emotional functioning: Week 96: number analyzed (Participants) | 3
  Emotional functioning: Week 96 | 11.11 (19.25)
  Emotional functioning: Week 99: number analyzed (Participants) | 1
  Emotional functioning: Week 99 | 0.00
  Emotional functioning: Week 105: number analyzed (Participants) | 1
  Emotional functioning: Week 105 | 0.00
  Emotional functioning: Week 111: number analyzed (Participants) | 1
  Emotional functioning: Week 111 | 0.00
  Emotional functioning: Week 117: number analyzed (Participants) | 1
  Emotional functioning: Week 117 | 0.00
  Emotional functioning: Last visit: number analyzed (Participants) | 73
  Emotional functioning: Last visit | 4.76 (19.86)
  Cognitive functioning: Baseline | 77.85 (24.13)
  Cognitive functioning: Week 6: number analyzed (Participants) | 64
  Cognitive functioning: Week 6 | 2.34 (20.76)
  Cognitive functioning: Week 9: number analyzed (Participants) | 1
  Cognitive functioning: Week 9 | 0.00
  Cognitive functioning: Week 12: number analyzed (Participants) | 54
  Cognitive functioning: Week 12 | 2.78 (15.44)
  Cognitive functioning: Week 15: number analyzed (Participants) | 1
  Cognitive functioning: Week 15 | 0.00
  Cognitive functioning: Week 18: number analyzed (Participants) | 49
  Cognitive functioning: Week 18 | 2.04 (15.82)
  Cognitive functioning: Week 21: number analyzed (Participants) | 1
  Cognitive functioning: Week 21 | 0.00
  Cognitive functioning: Week 24: number analyzed (Participants) | 41
  Cognitive functioning: Week 24 | -3.25 (16.34)
  Cognitive functioning: Week 27: number analyzed (Participants) | 2
  Cognitive functioning: Week 27 | 0.00 (0.00)
  Cognitive functioning: Week 30: number analyzed (Participants) | 39
  Cognitive functioning: Week 30 | -1.28 (17.68)
  Cognitive functioning: Week 33: number analyzed (Participants) | 3
  Cognitive functioning: Week 33 | -27.78 (25.46)
  Cognitive functioning: Week 36: number analyzed (Participants) | 38
  Cognitive functioning: Week 36 | -2.63 (13.16)
  Cognitive functioning: Week 39: number analyzed (Participants) | 2
  Cognitive functioning: Week 39 | -25.00 (35.36)
  Cognitive functioning: Week 42: number analyzed (Participants) | 36
  Cognitive functioning: Week 42 | -0.46 (14.08)
  Cognitive functioning Week 45: number analyzed (Participants) | 4
  Cognitive functioning Week 45 | -4.17 (51.59)
  Cognitive functioning: Week 48: number analyzed (Participants) | 33
  Cognitive functioning: Week 48 | -6.06 (21.58)
  Cognitive functioning: Week 51: number analyzed (Participants) | 2
  Cognitive functioning: Week 51 | -33.33 (0.00)
  Cognitive functioning: Week 54: number analyzed (Participants) | 31
  Cognitive functioning: Week 54 | -7.53 (22.29)
  Cognitive functioning: Week 57: number analyzed (Participants) | 5
  Cognitive functioning: Week 57 | 0.00 (31.18)
  Cognitive functioning: Week 60: number analyzed (Participants) | 30
  Cognitive functioning: Week 60 | -6.11 (21.66)
  Cognitive functioning: Week 63: number analyzed (Participants) | 3
  Cognitive functioning: Week 63 | 11.11 (19.25)
  Cognitive functioning: Week 66: number analyzed (Participants) | 26
  Cognitive functioning: Week 66 | -8.97 (22.23)
  Cognitive functioning: Week 69: number analyzed (Participants) | 4
  Cognitive functioning: Week 69 | 4.17 (8.33)
  Cognitive functioning: Week 72: number analyzed (Participants) | 23
  Cognitive functioning: Week 72 | -7.97 (20.64)
  Cognitive functioning: Week 75: number analyzed (Participants) | 2
  Cognitive functioning: Week 75 | 0.00 (0.00)
  Cognitive functioning: Week 78: number analyzed (Participants) | 21
  Cognitive functioning: Week 78 | -9.52 (25.59)
  Cognitive functioning: Week 81: number analyzed (Participants) | 2
  Cognitive functioning: Week 81 | 0.00 (0.00)
  Cognitive functioning: Week 84: number analyzed (Participants) | 13
  Cognitive functioning: Week 84 | -3.85 (20.59)
  Cognitive functioning: Week 87: number analyzed (Participants) | 3
  Cognitive functioning: Week 87 | -11.11 (19.25)
  Cognitive functioning: Week 90: number analyzed (Participants) | 8
  Cognitive functioning: Week 90 | -8.33 (15.43)
  Cognitive functioning: Week 93: number analyzed (Participants) | 2
  Cognitive functioning: Week 93 | 0.00 (0.00)
  Cognitive functioning: Week 96: number analyzed (Participants) | 3
  Cognitive functioning: Week 96 | -22.22 (19.25)
  Cognitive functioning: Week 99: number analyzed (Participants) | 1
  Cognitive functioning: Week 99 | 0.00
  Cognitive functioning: Week 105: number analyzed (Participants) | 1
  Cognitive functioning: Week 105 | 0.00
  Cognitive functioning: Week 111: number analyzed (Participants) | 1
  Cognitive functioning: Week 111 | 0.00
  Cognitive functioning: Week 117: number analyzed (Participants) | 1
  Cognitive functioning: Week 117 | 0.00
  Cognitive functioning: Last visit: number analyzed (Participants) | 73
  Cognitive functioning: Last visit | -4.79 (24.45)
  Social functioning: Baseline | 60.55 (35.32)
  Social functioning: Week 6: number analyzed (Participants) | 64
  Social functioning: Week 6 | 11.20 (23.20)
  Social functioning: Week 9: number analyzed (Participants) | 1
  Social functioning: Week 9 | 0.00
  Social functioning: Week 12: number analyzed (Participants) | 54
  Social functioning: Week 12 | 10.19 (27.93)
  Social functioning: Week 15: number analyzed (Participants) | 1
  Social functioning: Week 15 | 0.00
  Social functioning: Week 18: number analyzed (Participants) | 49
  Social functioning: Week 18 | 13.27 (25.45)
  Social functioning: Week 21: number analyzed (Participants) | 1
  Social functioning: Week 21 | 0.00
  Social functioning: Week 24: number analyzed (Participants) | 41
  Social functioning: Week 24 | 8.54 (26.38)
  Social functioning: Week 27: number analyzed (Participants) | 2
  Social functioning: Week 27 | 16.67 (23.57)
  Social functioning: Week 30: number analyzed (Participants) | 39
  Social functioning: Week 30 | 14.53 (31.11)
  Social functioning: Week 33: number analyzed (Participants) | 3
  Social functioning: Week 33 | 5.56 (25.46)
  Social functioning: Week 36: number analyzed (Participants) | 38
  Social functioning: Week 36 | 9.21 (32.35)
  Social functioning: Week 39: number analyzed (Participants) | 2
  Social functioning: Week 39 | -8.33 (11.79)
  Social functioning: Week 42: number analyzed (Participants) | 36
  Social functioning: Week 42 | 8.80 (30.47)
  Social functioning: Week 45: number analyzed (Participants) | 4
  Social functioning: Week 45 | 4.17 (20.97)
  Social functioning: Week 48: number analyzed (Participants) | 33
  Social functioning: Week 48 | 16.16 (29.31)
  Social functioning: Week 51: number analyzed (Participants) | 2
  Social functioning: Week 51 | -8.33 (11.79)
  Social functioning: Week 54: number analyzed (Participants) | 31
  Social functioning: Week 54 | 12.37 (28.53)
  Social functioning: Week 57: number analyzed (Participants) | 5
  Social functioning: Week 57 | 3.33 (18.26)
  Social functioning: Week 60: number analyzed (Participants) | 30
  Social functioning: Week 60 | 8.33 (25.43)
  Social functioning: Week 63: number analyzed (Participants) | 3
  Social functioning: Week 63 | 0.00 (33.33)
  Social functioning: Week 66: number analyzed (Participants) | 26
  Social functioning: Week 66 | 5.77 (31.95)
  Social functioning: Week 69: number analyzed (Participants) | 4
  Social functioning: Week 69 | 20.83 (25.00)
  Social functioning: Week 72: number analyzed (Participants) | 23
  Social functioning: Week 72 | 11.59 (23.80)
  Social functioning: Week 75: number analyzed (Participants) | 2
  Social functioning: Week 75 | 16.67 (23.57)
  Social functioning: Week 78: number analyzed (Participants) | 21
  Social functioning: Week 78 | 12.70 (23.51)
  Social functioning: Week 81: number analyzed (Participants) | 2
  Social functioning: Week 81 | 16.67 (23.57)
  Social functioning: Week 84: number analyzed (Participants) | 13
  Social functioning: Week 84 | 8.97 (29.36)
  Social functioning: Week 87: number analyzed (Participants) | 3
  Social functioning: Week 87 | 27.78 (25.46)
  Social functioning: Week 90: number analyzed (Participants) | 8
  Social functioning: Week 90 | 14.58 (16.52)
  Social functioning: Week 93: number analyzed (Participants) | 2
  Social functioning: Week 93 | -8.33 (82.50)
  Social functioning: Week 96: number analyzed (Participants) | 3
  Social functioning: Week 96 | 16.67 (16.67)
  Social functioning: Week 99: number analyzed (Participants) | 1
  Social functioning: Week 99 | 0.00
  Social functioning: Week 105: number analyzed (Participants) | 1
  Social functioning: Week 105 | 0.00
  Social functioning: Week 111: number analyzed (Participants) | 1
  Social functioning: Week 111 | 0.00
  Social functioning: Week 117: number analyzed (Participants) | 1
  Social functioning: Week 117 | 0.00
  Social functioning: Last visit: number analyzed (Participants) | 73
  Social functioning: Last visit | 3.20 (30.39)
  Fatigue: Baseline | 45.57 (27.02)
  Fatigue: Week 6: number analyzed (Participants) | 64
  Fatigue: Week 6 | -10.94 (25.70)
  Fatigue: Week 9: number analyzed (Participants) | 1
  Fatigue: Week 9 | -11.11
  Fatigue: Week 12: number analyzed (Participants) | 54
  Fatigue: Week 12 | -11.11 (27.73)
  Fatigue: Week 15: number analyzed (Participants) | 1
  Fatigue: Week 15 | 0.00
  Fatigue: Week 18: number analyzed (Participants) | 51
  Fatigue: Week 18 | -12.85 (24.88)
  Fatigue: Week 21: number analyzed (Participants) | 1
  Fatigue: Week 21 | 0.00
  Fatigue: Week 24: number analyzed (Participants) | 42
  Fatigue: Week 24 | -10.05 (22.06)
  Fatigue: Week 27: number analyzed (Participants) | 2
  Fatigue: Week 27 | 5.56 (7.86)
  Fatigue: Week 30: number analyzed (Participants) | 39
  Fatigue: Week 30 | -9.97 (23.47)
  Fatigue: Week 33: number analyzed (Participants) | 3
  Fatigue: Week 33 | 14.81 (6.42)
  Fatigue: Week 36: number analyzed (Participants) | 38
  Fatigue: Week 36 | -10.23 (25.75)
  Fatigue: Week 39: number analyzed (Participants) | 2
  Fatigue: Week 39 | 5.56 (7.86)
  Fatigue: Week 42: number analyzed (Participants) | 36
  Fatigue: Week 42 | -9.26 (21.50)
  Fatigue: Week 45: number analyzed (Participants) | 4
  Fatigue: Week 45 | 0.00 (24.00)
  Fatigue: Week 48: number analyzed (Participants) | 32
  Fatigue: Week 48 | -11.11 (22.93)
  Fatigue: Week 51: number analyzed (Participants) | 2
  Fatigue: Week 51 | 0.00 (47.14)
  Fatigue: Week 54: number analyzed (Participants) | 32
  Fatigue: Week 54 | -7.64 (18.39)
  Fatigue: Week 57: number analyzed (Participants) | 5
  Fatigue: Week 57 | 4.44 (16.85)
  Fatigue: Week 60: number analyzed (Participants) | 30
  Fatigue: Week 60 | -7.78 (21.27)
  Fatigue: Week 63: number analyzed (Participants) | 3
  Fatigue: Week 63 | 7.41 (23.13)
  Fatigue: Week 66: number analyzed (Participants) | 26
  Fatigue: Week 66 | -7.69 (20.07)
  Fatigue: Week 69: number analyzed (Participants) | 4
  Fatigue: Week 69 | -8.33 (10.64)
  Fatigue: Week 72: number analyzed (Participants) | 23
  Fatigue: Week 72 | -8.21 (22.28)
  Fatigue: Week 75: number analyzed (Participants) | 2
  Fatigue: Week 75 | -5.56 (7.86)
  Fatigue: Week 78: number analyzed (Participants) | 21
  Fatigue: Week 78 | -6.35 (23.19)
  Fatigue: Week 81: number analyzed (Participants) | 2
  Fatigue: Week 81 | -5.56 (7.86)
  Fatigue: Week 84: number analyzed (Participants) | 13
  Fatigue: Week 84 | -9.40 (18.62)
  Fatigue: Week 87: number analyzed (Participants) | 3
  Fatigue: Week 87 | 0.00 (11.11)
  Fatigue: Week 90: number analyzed (Participants) | 8
  Fatigue: Week 90 | -8.33 (17.57)
  Fatigue: Week 93: number analyzed (Participants) | 2
  Fatigue: Week 93 | 33.33 (31.43)
  Fatigue: Week 96: number analyzed (Participants) | 3
  Fatigue: Week 96 | -18.52 (6.42)
  Fatigue: Week 99: number analyzed (Participants) | 1
  Fatigue: Week 99 | 0.00
  Fatigue: Week 105: number analyzed (Participants) | 1
  Fatigue: Week 105 | 0.00
  Fatigue: Week 111: number analyzed (Participants) | 1
  Fatigue: Week 111 | 0.00
  Fatigue: Week 117: number analyzed (Participants) | 1
  Fatigue: Week 117 | 0.00
  Fatigue: Last visit: number analyzed (Participants) | 73
  Fatigue: Last visit | -6.85 (21.65)
  Nausea and vomiting: Baseline | 15.61 (20.73)
  Nausea and vomiting: Week 6: number analyzed (Participants) | 64
  Nausea and vomiting: Week 6 | -6.77 (19.63)
  Nausea and vomiting: Week 9: number analyzed (Participants) | 1
  Nausea and vomiting: Week 9 | 0.00
  Nausea and vomiting: Week 12: number analyzed (Participants) | 54
  Nausea and vomiting: Week 12 | -8.02 (21.66)
  Nausea and vomiting: Week 15: number analyzed (Participants) | 1
  Nausea and vomiting: Week 15 | 0.00
  Nausea and vomiting: Week 18: number analyzed (Participants) | 51
  Nausea and vomiting: Week 18 | -9.15 (19.81)
  Nausea and vomiting: Week 21: number analyzed (Participants) | 1
  Nausea and vomiting: Week 21 | 0.00
  Nausea and vomiting: Week 24: number analyzed (Participants) | 42
  Nausea and vomiting: Week 24 | -9.13 (18.48)
  Nausea and vomiting: Week 27: number analyzed (Participants) | 2
  Nausea and vomiting: Week 27 | -8.33 (11.79)
  Nausea and vomiting: Week 30: number analyzed (Participants) | 39
  Nausea and vomiting: Week 30 | -5.98 (17.31)
  Nausea and vomiting: Week 33: number analyzed (Participants) | 3
  Nausea and vomiting: Week 33 | 11.11 (25.46)
  Nausea and vomiting: Week 36: number analyzed (Participants) | 38
  Nausea and vomiting: Week 36 | -7.46 (17.63)
  Nausea and vomiting: Week 39: number analyzed (Participants) | 2
  Nausea and vomiting: Week 39 | 16.67 (23.57)
  Nausea and vomiting: Week 42: number analyzed (Participants) | 36
  Nausea and vomiting: Week 42 | -8.80 (18.47)
  Nausea and vomiting: Week 45: number analyzed (Participants) | 4
  Nausea and vomiting: Week 45 | 4.17 (8.33)
  Nausea and vomiting: Week 48: number analyzed (Participants) | 32
  Nausea and vomiting: Week 48 | -9.38 (19.37)
  Nausea and vomiting: Week 51: number analyzed (Participants) | 2
  Nausea and vomiting: Week 51 | 8.33 (11.79)
  Nausea and vomiting: Week 54: number analyzed (Participants) | 32
  Nausea and vomiting: Week 54 | -8.85 (19.85)
  Nausea and vomiting: Week 57: number analyzed (Participants) | 5
  Nausea and vomiting: Week 57 | 6.67 (14.91)
  Nausea and vomiting: Week 60: number analyzed (Participants) | 30
  Nausea and vomiting: Week 60 | -6.67 (17.29)
  Nausea and vomiting: Week 63: number analyzed (Participants) | 3
  Nausea and vomiting: Week 63 | 11.11 (19.25)
  Nausea and vomiting: Week 66: number analyzed (Participants) | 26
  Nausea and vomiting: Week 66 | -7.05 (20.10)
  Nausea and vomiting: Week 69: number analyzed (Participants) | 4
  Nausea and vomiting: Week 69 | 0.00 (0.00)
  Nausea and vomiting: Week 72: number analyzed (Participants) | 23
  Nausea and vomiting: Week 72 | -5.80 (19.85)
  Nausea and vomiting: Week 75: number analyzed (Participants) | 2
  Nausea and vomiting: Week 75 | 0.00 (0.00)
  Nausea and vomiting: Week 78: number analyzed (Participants) | 21
  Nausea and vomiting: Week 78 | -5.56 (13.26)
  Nausea and vomiting: Week 81: number analyzed (Participants) | 2
  Nausea and vomiting: Week 81 | 0.00 (0.00)
  Nausea and vomiting: Week 84: number analyzed (Participants) | 13
  Nausea and vomiting: Week 84 | -6.41 (12.80)
  Nausea and vomiting: Week 87: number analyzed (Participants) | 3
  Nausea and vomiting: Week 87 | 5.56 (9.62)
  Nausea and vomiting: Week 90: number analyzed (Participants) | 8
  Nausea and vomiting: Week 90 | 2.08 (13.91)
  Nausea and vomiting: Week 93: number analyzed (Participants) | 2
  Nausea and vomiting: Week 93 | 0.00 (0.00)
  Nausea and vomiting: Week 96: number analyzed (Participants) | 3
  Nausea and vomiting: Week 96 | 0.00 (16.67)
  Nausea and vomiting: Week 99: number analyzed (Participants) | 1
  Nausea and vomiting: Week 99 | 0.00
  Nausea and vomiting: Week 105: number analyzed (Participants) | 1
  Nausea and vomiting: Week 105 | 0.00
  Nausea and vomiting: Week 111: number analyzed (Participants) | 1
  Nausea and vomiting: Week 111 | 0.00
  Nausea and vomiting: Week 117: number analyzed (Participants) | 1
  Nausea and vomiting: Week 117 | 0.00
  Nausea and vomiting: Last visit: number analyzed (Participants) | 73
  Nausea and vomiting: Last visit | -6.85 (20.38)
  Pain: Baseline | 36.29 (33.63)
  Pain: Week 6: number analyzed (Participants) | 64
  Pain: Week 6 | -12.50 (33.47)
  Pain: Week 9: number analyzed (Participants) | 1
  Pain: Week 9 | 0.00
  Pain: Week 12: number analyzed (Participants) | 54
  Pain: Week 12 | -14.81 (32.48)
  Pain: Week 15: number analyzed (Participants) | 1
  Pain: Week 15 | 0.00
  Pain: Week 18: number analyzed (Participants) | 51
  Pain: Week 18 | -13.07 (33.55)
  Pain: Week 21: number analyzed (Participants) | 1
  Pain: Week 21 | 0.00
  Pain: Week 24: number analyzed (Participants) | 42
  Pain: Week 24 | -6.35 (31.44)
  Pain: Week 27: number analyzed (Participants) | 2
  Pain: Week 27 | 8.33 (11.79)
  Pain: Week 30: number analyzed (Participants) | 39
  Pain: Week 30 | -5.13 (33.37)
  Pain: Week 33: number analyzed (Participants) | 3
  Pain: Week 33 | 5.56 (9.62)
  Pain: Week 36: number analyzed (Participants) | 38
  Pain: Week 36 | -6.14 (34.31)
  Pain: Week 39: number analyzed (Participants) | 2
  Pain: Week 39 | -8.33 (11.79)
  Pain: Week 42: number analyzed (Participants) | 36
  Pain: Week 42 | -5.09 (23.17)
  Pain: Week 45: number analyzed (Participants) | 4
  Pain: Week 45 | 8.33 (21.52)
  Pain: Week 48: number analyzed (Participants) | 33
  Pain: Week 48 | -4.55 (17.81)
  Pain: Week 51: number analyzed (Participants) | 2
  Pain: Week 51 | -25.00 (11.79)
  Pain: Week 54: number analyzed (Participants) | 32
  Pain: Week 54 | -0.52 (24.86)
  Pain: Week 57: number analyzed (Participants) | 5
  Pain: Week 57 | 0.00 (39.09)
  Pain: Week 60: number analyzed (Participants) | 30
  Pain: Week 60 | 0.56 (14.17)
  Pain: Week 63: number analyzed (Participants) | 3
  Pain: Week 63 | -5.56 (9.62)
  Pain: Week 66: number analyzed (Participants) | 26
  Pain: Week 66 | -5.13 (23.46)
  Pain: Week 69: number analyzed (Participants) | 4
  Pain: Week 69 | -4.17 (15.96)
  Pain: Week 72: number analyzed (Participants) | 23
  Pain: Week 72 | -5.07 (28.62)
  Pain: Week 75: number analyzed (Participants) | 2
  Pain: Week 75 | -8.33 (11.79)
  Pain: Week 78: number analyzed (Participants) | 21
  Pain: Week 78 | 1.59 (15.73)
  Pain: Week 81: number analyzed (Participants) | 2
  Pain: Week 81 | -8.33 (11.79)
  Pain: Week 84: number analyzed (Participants) | 13
  Pain: Week 84 | -5.13 (19.70)
  Pain: Week 87: number analyzed (Participants) | 3
  Pain: Week 87 | -5.56 (9.62)
  Pain: Week 90: number analyzed (Participants) | 8
  Pain: Week 90 | -8.33 (25.20)
  Pain: Week 93: number analyzed (Participants) | 2
  Pain: Week 93 | 25.00 (35.36)
  Pain: Week 96: number analyzed (Participants) | 3
  Pain: Week 96 | -11.11 (53.58)
  Pain: Week 99: number analyzed (Participants) | 1
  Pain: Week 99 | 0.00
  Pain: Week 105: number analyzed (Participants) | 1
  Pain: Week 105 | 0.00
  Pain: Week 111: number analyzed (Participants) | 1
  Pain: Week 111 | 0.00
  Pain: Week 117: number analyzed (Participants) | 1
  Pain: Week 117 | 0.00
  Pain: Last visit: number analyzed (Participants) | 73
  Pain: Last visit | -9.36 (29.92)
  Dyspnoea: Baseline: number analyzed (Participants) | 78
  Dyspnoea: Baseline | 33.33 (30.86)
  Dyspnoea: Week 6: number analyzed (Participants) | 63
  Dyspnoea: Week 6 | -12.17 (32.96)
  Dyspnoea : Week 9: number analyzed (Participants) | 1
  Dyspnoea : Week 9 | 0.00
  Dyspnoea: Week 12: number analyzed (Participants) | 53
  Dyspnoea: Week 12 | -10.69 (32.54)
  Dyspnoea: Week 15: number analyzed (Participants) | 1
  Dyspnoea: Week 15 | 0.00
  Dyspnoea: Week 18: number analyzed (Participants) | 50
  Dyspnoea: Week 18 | -12.67 (30.78)
  Dyspnoea: Week 21: number analyzed (Participants) | 1
  Dyspnoea: Week 21 | 0.00
  Dyspnoea: Week 24: number analyzed (Participants) | 40
  Dyspnoea: Week 24 | -7.50 (25.58)
  Dyspnoea: Week 27: number analyzed (Participants) | 2
  Dyspnoea: Week 27 | 0.00 (0.00)
  Dyspnoea: Week 30: number analyzed (Participants) | 38
  Dyspnoea: Week 30 | -7.89 (26.21)
  Dyspnoea: Week 33: number analyzed (Participants) | 3
  Dyspnoea: Week 33 | 0.00 (33.33)
  Dyspnoea: Week 36: number analyzed (Participants) | 37
  Dyspnoea: Week 36 | -7.21 (27.37)
  Dyspnoea: Week 39: number analyzed (Participants) | 2
  Dyspnoea: Week 39 | -16.67 (23.57)
  Dyspnoea: Week 42: number analyzed (Participants) | 35
  Dyspnoea: Week 42 | -5.71 (27.40)
  Dyspnoea: Week 45: number analyzed (Participants) | 4
  Dyspnoea: Week 45 | 0.00 (27.22)
  Dyspnoea: Week 48: number analyzed (Participants) | 32
  Dyspnoea: Week 48 | -6.25 (28.63)
  Dyspnoea: Week 51: number analyzed (Participants) | 2
  Dyspnoea: Week 51 | 0.00 (0.00)
  Dyspnoea: Week 54: number analyzed (Participants) | 32
  Dyspnoea: Week 54 | -7.29 (23.55)
  Dyspnoea: Week 57: number analyzed (Participants) | 5
  Dyspnoea: Week 57 | -6.67 (14.91)
  Dyspnoea: Week 60: number analyzed (Participants) | 30
  Dyspnoea: Week 60 | -1.11 (22.29)
  Dyspnoea: Week 63: number analyzed (Participants) | 3
  Dyspnoea: Week 63 | -11.11 (19.25)
  Dyspnoea: Week 66: number analyzed (Participants) | 26
  Dyspnoea: Week 66 | -8.97 (24.14)
  Dyspnoea: Week 69: number analyzed (Participants) | 4
  Dyspnoea: Week 69 | -8.33 (16.67)
  Dyspnoea: Week 72: number analyzed (Participants) | 23
  Dyspnoea: Week 72 | -1.45 (32.53)
  Dyspnoea: Week 75: number analyzed (Participants) | 2
  Dyspnoea: Week 75 | -16.67 (23.57)
  Dyspnoea: Week 78: number analyzed (Participants) | 21
  Dyspnoea: Week 78 | -4.76 (21.82)
  Dyspnoea: Week 81: number analyzed (Participants) | 2
  Dyspnoea: Week 81 | -16.67 (23.57)
  Dyspnoea: Week 84: number analyzed (Participants) | 13
  Dyspnoea: Week 84 | 0.00 (23.57)
  Dyspnoea: Week 87: number analyzed (Participants) | 3
  Dyspnoea: Week 87 | -11.11 (19.25)
  Dyspnoea: Week 90: number analyzed (Participants) | 8
  Dyspnoea: Week 90 | 8.33 (29.55)
  Dyspnoea: Week 93: number analyzed (Participants) | 2
  Dyspnoea: Week 93 | 16.67 (23.57)
  Dyspnoea: Week 96: number analyzed (Participants) | 3
  Dyspnoea: Week 96 | -11.11 (38.49)
  Dyspnoea: Week 99: number analyzed (Participants) | 1
  Dyspnoea: Week 99 | 33.33
  Dyspnoea: Week 105: number analyzed (Participants) | 1
  Dyspnoea: Week 105 | 0.00
  Dyspnoea: Week 111: number analyzed (Participants) | 1
  Dyspnoea: Week 111 | 0.00
  Dyspnoea: Week 117: number analyzed (Participants) | 1
  Dyspnoea: Week 117 | 0.00
  Dyspnoea: Last visit: number analyzed (Participants) | 72
  Dyspnoea: Last visit | -4.63 (33.71)
  Insomnia: Baseline | 31.22 (30.82)
  Insomnia: Week 6: number analyzed (Participants) | 64
  Insomnia: Week 6 | -9.38 (29.38)
  Insomnia: Week 9: number analyzed (Participants) | 1
  Insomnia: Week 9 | 0.00
  Insomnia: Week 12: number analyzed (Participants) | 54
  Insomnia: Week 12 | -9.26 (34.52)
  Insomnia: Week 15: number analyzed (Participants) | 1
  Insomnia: Week 15 | 0.00
  Insomnia: Week 18: number analyzed (Participants) | 51
  Insomnia: Week 18 | -3.27 (37.86)
  Insomnia: Week 21: number analyzed (Participants) | 1
  Insomnia: Week 21 | 0.00
  Insomnia: Week 24: number analyzed (Participants) | 42
  Insomnia: Week 24 | -3.17 (36.67)
  Insomnia: Week 27: number analyzed (Participants) | 2
  Insomnia: Week 27 | 0.00 (0.00)
  Insomnia: Week 30: number analyzed (Participants) | 39
  Insomnia: Week 30 | -9.40 (33.29)
  Insomnia: Week 33: number analyzed (Participants) | 3
  Insomnia: Week 33 | 44.44 (50.92)
  Insomnia: Week 36: number analyzed (Participants) | 38
  Insomnia: Week 36 | -8.77 (40.03)
  Insomnia: Week 39: number analyzed (Participants) | 2
  Insomnia: Week 39 | 83.33 (23.57)
  Insomnia: Week 42: number analyzed (Participants) | 36
  Insomnia: Week 42 | -5.56 (25.82)
  Insomnia: Week 45: number analyzed (Participants) | 4
  Insomnia: Week 45 | 41.67 (31.91)
  Insomnia: Week 48: number analyzed (Participants) | 32
  Insomnia: Week 48 | -3.13 (29.77)
  Insomnia: Week 51: number analyzed (Participants) | 2
  Insomnia: Week 51 | 50.00 (23.57)
  Insomnia: Week 54: number analyzed (Participants) | 32
  Insomnia: Week 54 | -2.08 (28.00)
  Insomnia: Week 57: number analyzed (Participants) | 5
  Insomnia: Week 57 | 40.00 (43.46)
  Insomnia: Week 60: number analyzed (Participants) | 30
  Insomnia: Week 60 | -1.11 (28.34)
  Insomnia: Week 63: number analyzed (Participants) | 3
  Insomnia: Week 63 | 0.00 (33.33)
  Insomnia: Week 66: number analyzed (Participants) | 25
  Insomnia: Week 66 | -5.33 (32.89)
  Insomnia: Week 69: number analyzed (Participants) | 4
  Insomnia: Week 69 | 0.00 (27.22)
  Insomnia: Week 72: number analyzed (Participants) | 23
  Insomnia: Week 72 | 0.00 (26.59)
  Insomnia: Week 75: number analyzed (Participants) | 2
  Insomnia: Week 75 | 0.00 (0.00)
  Insomnia: Week 78: number analyzed (Participants) | 21
  Insomnia: Week 78 | 1.59 (22.30)
  Insomnia: Week 81: number analyzed (Participants) | 2
  Insomnia: Week 81 | 0.00 (0.00)
  Insomnia: Week 84: number analyzed (Participants) | 13
  Insomnia: Week 84 | 0.00 (36.00)
  Insomnia: Week 87: number analyzed (Participants) | 3
  Insomnia: Week 87 | 11.11 (19.25)
  Insomnia: Week 90: number analyzed (Participants) | 8
  Insomnia: Week 90 | 0.00 (30.86)
  Insomnia: Week 93: number analyzed (Participants) | 2
  Insomnia: Week 93 | 0.00 (0.00)
  Insomnia: Week 96: number analyzed (Participants) | 3
  Insomnia: Week 96 | 22.22 (38.49)
  Insomnia: Week 99: number analyzed (Participants) | 1
  Insomnia: Week 99 | 0.00
  Insomnia: Week 105: number analyzed (Participants) | 1
  Insomnia: Week 105 | 0.00
  Insomnia: Week 111: number analyzed (Participants) | 1
  Insomnia: Week 111 | 0.00
  Insomnia: Week 117: number analyzed (Participants) | 1
  Insomnia: Week 117 | 0.00
  Insomnia: Last visit: number analyzed (Participants) | 73
  Insomnia: Last visit | -1.83 (35.09)
  Appetite loss: Baseline | 29.96 (33.16)
  Appetite loss: Week 6: number analyzed (Participants) | 64
  Appetite loss: Week 6 | -16.67 (30.28)
  Appetite loss: Week 9: number analyzed (Participants) | 1
  Appetite loss: Week 9 | 0.00
  Appetite loss: Week 12: number analyzed (Participants) | 54
  Appetite loss: Week 12 | -18.52 (36.44)
  Appetite loss: Week 15: number analyzed (Participants) | 1
  Appetite loss: Week 15 | 0.00
  Appetite loss: Week 18: number analyzed (Participants) | 51
  Appetite loss: Week 18 | -20.26 (33.39)
  Appetite loss: Week 21: number analyzed (Participants) | 1
  Appetite loss: Week 21 | 0.00
  Appetite loss: Week 24: number analyzed (Participants) | 42
  Appetite loss: Week 24 | -19.84 (29.50)
  Appetite loss: Week 27: number analyzed (Participants) | 2
  Appetite loss: Week 27 | -16.67 (23.57)
  Appetite loss: Week 30: number analyzed (Participants) | 39
  Appetite loss: Week 30 | -13.68 (23.84)
  Appetite loss: Week 33: number analyzed (Participants) | 3
  Appetite loss: Week 33 | -44.44 (19.25)
  Appetite loss: Week 36: number analyzed (Participants) | 38
  Appetite loss: Week 36 | -14.91 (27.62)
  Appetite loss: Week 39: number analyzed (Participants) | 2
  Appetite loss: Week 39 | -50.00 (23.57)
  Appetite loss: Week 42: number analyzed (Participants) | 36
  Appetite loss: Week 42 | -16.67 (32.37)
  Appetite loss: Week 45: number analyzed (Participants) | 4
  Appetite loss: Week 45 | -8.33 (41.94)
  Appetite loss: Week 48: number analyzed (Participants) | 32
  Appetite loss: Week 48 | -20.83 (34.65)
  Appetite loss: Week 51: number analyzed (Participants) | 2
  Appetite loss: Week 51 | -33.33 (47.14)
  Appetite loss: Week 54: number analyzed (Participants) | 32
  Appetite loss: Week 54 | -18.75 (32.72)
  Appetite loss: Week 57: number analyzed (Participants) | 5
  Appetite loss: Week 57 | -20.00 (29.81)
  Appetite loss: Week 60: number analyzed (Participants) | 30
  Appetite loss: Week 60 | -20.00 (31.07)
  Appetite loss: Week 63: number analyzed (Participants) | 3
  Appetite loss: Week 63 | 0.00 (0.00)
  Appetite loss: Week 66: number analyzed (Participants) | 26
  Appetite loss: Week 66 | -23.08 (33.69)
  Appetite loss: Week 69: number analyzed (Participants) | 4
  Appetite loss: Week 69 | -16.67 (33.33)
  Appetite loss: Week 72: number analyzed (Participants) | 23
  Appetite loss: Week 72 | -23.19 (30.87)
  Appetite loss: Week 75: number analyzed (Participants) | 2
  Appetite loss: Week 75 | 0.00 (0.00)
  Appetite loss: Week 78: number analyzed (Participants) | 21
  Appetite loss: Week 78 | -20.63 (30.69)
  Appetite loss: Week 81: number analyzed (Participants) | 2
  Appetite loss: Week 81 | 0.00 (0.00)
  Appetite loss: Week 84: number analyzed (Participants) | 13
  Appetite loss: Week 84 | -25.64 (36.40)
  Appetite loss: Week 87: number analyzed (Participants) | 3
  Appetite loss: Week 87 | 11.11 (19.25)
  Appetite loss: Week 90: number analyzed (Participants) | 8
  Appetite loss: Week 90 | -20.83 (39.59)
  Appetite loss: Week 93: number analyzed (Participants) | 2
  Appetite loss: Week 93 | 0.00 (0.00)
  Appetite loss: Week 96: number analyzed (Participants) | 3
  Appetite loss: Week 96 | -55.56 (50.92)
  Appetite loss: Week 99: number analyzed (Participants) | 1
  Appetite loss: Week 99 | 0.00
  Appetite loss: Week 105: number analyzed (Participants) | 1
  Appetite loss: Week 105 | 0.00
  Appetite loss: Week 111: number analyzed (Participants) | 1
  Appetite loss: Week 111 | 0.00
  Appetite loss: Week 117: number analyzed (Participants) | 1
  Appetite loss: Week 117 | 0.00
  Appetite loss: Last visit: number analyzed (Participants) | 73
  Appetite loss: Last visit | -13.70 (33.72)
  Constipation: Baseline | 20.25 (26.38)
  Constipation: Week 6: number analyzed (Participants) | 64
  Constipation: Week 6 | 9.90 (30.68)
  Constipation: Week 9: number analyzed (Participants) | 1
  Constipation: Week 9 | 0.00
  Constipation: Week 12: number analyzed (Participants) | 54
  Constipation: Week 12 | 1.85 (31.33)
  Constipation: Week 15: number analyzed (Participants) | 1
  Constipation: Week 15 | 33.33
  Constipation: Week 18: number analyzed (Participants) | 51
  Constipation: Week 18 | 4.58 (25.84)
  Constipation: Week 21: number analyzed (Participants) | 1
  Constipation: Week 21 | 0.00
  Constipation: Week 24: number analyzed (Participants) | 42
  Constipation: Week 24 | 2.38 (29.81)
  Constipation: Week 27: number analyzed (Participants) | 2
  Constipation: Week 27 | 33.33 (47.14)
  Constipation: Week 30: number analyzed (Participants) | 39
  Constipation: Week 30 | 5.13 (27.08)
  Constipation: Week 33: number analyzed (Participants) | 3
  Constipation: Week 33 | 11.11 (50.92)
  Constipation: Week 36: number analyzed (Participants) | 38
  Constipation: Week 36 | 5.26 (21.26)
  Constipation: Week 39: number analyzed (Participants) | 2
  Constipation: Week 39 | 16.67 (23.57)
  Constipation: Week 42: number analyzed (Participants) | 36
  Constipation: Week 42 | 9.26 (24.70)
  Constipation: Week 45: number analyzed (Participants) | 4
  Constipation: Week 45 | 50.00 (19.25)
  Constipation: Week 48: number analyzed (Participants) | 32
  Constipation: Week 48 | 1.04 (26.07)
  Constipation: Week 51: number analyzed (Participants) | 2
  Constipation: Week 51 | -16.67 (23.57)
  Constipation: Week 54: number analyzed (Participants) | 31
  Constipation: Week 54 | 6.45 (23.44)
  Constipation: Week 57: number analyzed (Participants) | 5
  Constipation: Week 57 | 26.67 (43.46)
  Constipation: Week 60: number analyzed (Participants) | 30
  Constipation: Week 60 | 6.67 (22.15)
  Constipation: Week 63: number analyzed (Participants) | 3
  Constipation: Week 63 | 44.44 (38.49)
  Constipation: Week 66: number analyzed (Participants) | 26
  Constipation: Week 66 | 12.82 (26.79)
  Constipation: Week 69: number analyzed (Participants) | 4
  Constipation: Week 69 | -8.33 (16.67)
  Constipation: Week 72: number analyzed (Participants) | 23
  Constipation: Week 72 | 4.35 (25.23)
  Constipation: Week 75: number analyzed (Participants) | 2
  Constipation: Week 75 | 33.33 (47.14)
  Constipation: Week 78: number analyzed (Participants) | 21
  Constipation: Week 78 | 7.94 (17.97)
  Constipation: Week 81: number analyzed (Participants) | 2
  Constipation: Week 81 | 33.33 (47.14)
  Constipation: Week 84: number analyzed (Participants) | 13
  Constipation: Week 84 | 7.69 (19.97)
  Constipation: Week 87: number analyzed (Participants) | 3
  Constipation: Week 87 | 22.22 (38.49)
  Constipation: Week 90: number analyzed (Participants) | 8
  Constipation: Week 90 | 8.33 (15.43)
  Constipation: Week 93: number analyzed (Participants) | 2
  Constipation: Week 93 | 33.33 (47.14)
  Constipation: Week 96: number analyzed (Participants) | 3
  Constipation: Week 96 | -11.11 (50.92)
  Constipation: Week 99: number analyzed (Participants) | 1
  Constipation: Week 99 | 33.33
  Constipation: Week 105: number analyzed (Participants) | 1
  Constipation: Week 105 | 0.00
  Constipation: Week 111: number analyzed (Participants) | 1
  Constipation: Week 111 | 0.00
  Constipation: Week 117: number analyzed (Participants) | 1
  Constipation: Week 117 | 0.00
  Constipation: Last visit: number analyzed (Participants) | 73
  Constipation: Last visit | 8.68 (31.93)
  Diarrhoea: Baseline: number analyzed (Participants) | 78
  Diarrhoea: Baseline | 13.25 (23.01)
  Diarrhoea: Week 6: number analyzed (Participants) | 63
  Diarrhoea: Week 6 | -7.41 (25.00)
  Diarrhoea: Week 9: number analyzed (Participants) | 1
  Diarrhoea: Week 9 | 0.00
  Diarrhoea: Week 12: number analyzed (Participants) | 53
  Diarrhoea: Week 12 | -6.29 (23.62)
  Diarrhoea: Week 15: number analyzed (Participants) | 1
  Diarrhoea: Week 15 | 0.00
  Diarrhoea: Week 18: number analyzed (Participants) | 48
  Diarrhoea: Week 18 | -5.56 (25.11)
  Diarrhoea: Week 21: number analyzed (Participants) | 1
  Diarrhoea: Week 21 | 0.00
  Diarrhoea: Week 24: number analyzed (Participants) | 40
  Diarrhoea: Week 24 | -4.17 (28.43)
  Diarrhoea: Week 27: number analyzed (Participants) | 2
  Diarrhoea: Week 27 | -16.67 (23.57)
  Diarrhoea: Week 30: number analyzed (Participants) | 39
  Diarrhoea: Week 30 | -8.55 (23.84)
  Diarrhoea: Week 33: number analyzed (Participants) | 2
  Diarrhoea: Week 33 | -16.67 (23.57)
  Diarrhoea: Week 36: number analyzed (Participants) | 38
  Diarrhoea: Week 36 | -7.89 (23.80)
  Diarrhoea: Week 39: number analyzed (Participants) | 1
  Diarrhoea: Week 39 | 0.00
  Diarrhoea: Week 42: number analyzed (Participants) | 36
  Diarrhoea: Week 42 | -6.48 (26.21)
  Diarrhoea: Week 45: number analyzed (Participants) | 3
  Diarrhoea: Week 45 | 0.00 (0.00)
  Diarrhoea: Week 48: number analyzed (Participants) | 33
  Diarrhoea: Week 48 | -3.03 (28.09)
  Diarrhoea: Week 51: number analyzed (Participants) | 1
  Diarrhoea: Week 51 | 0.00
  Diarrhoea: Week 54: number analyzed (Participants) | 32
  Diarrhoea: Week 54 | -6.25 (26.01)
  Diarrhoea: Week 57: number analyzed (Participants) | 4
  Diarrhoea: Week 57 | 0.00 (0.00)
  Diarrhoea: Week 60: number analyzed (Participants) | 30
  Diarrhoea: Week 60 | -1.11 (32.14)
  Diarrhoea: Week 63: number analyzed (Participants) | 3
  Diarrhoea: Week 63 | 0.00 (0.00)
  Diarrhoea: Week 66: number analyzed (Participants) | 26
  Diarrhoea: Week 66 | -7.69 (30.27)
  Diarrhoea: Week 69: number analyzed (Participants) | 3
  Diarrhoea: Week 69 | 11.11 (19.25)
  Diarrhoea: Week 72: number analyzed (Participants) | 23
  Diarrhoea: Week 72 | -7.25 (28.35)
  Diarrhoea: Week 75: number analyzed (Participants) | 2
  Diarrhoea: Week 75 | 0.00 (0.00)
  Diarrhoea: Week 78: number analyzed (Participants) | 20
  Diarrhoea: Week 78 | -6.67 (25.59)
  Diarrhoea: Week 81: number analyzed (Participants) | 2
  Diarrhoea: Week 81 | 0.00 (0.00)
  Diarrhoea: Week 84: number analyzed (Participants) | 12
  Diarrhoea: Week 84 | 2.78 (26.43)
  Diarrhoea: Week 87: number analyzed (Participants) | 3
  Diarrhoea: Week 87 | 11.11 (19.25)
  Diarrhoea: Week 90: number analyzed (Participants) | 7
  Diarrhoea: Week 90 | 9.52 (16.27)
  Diarrhoea: Week 93: number analyzed (Participants) | 2
  Diarrhoea: Week 93 | 0.00 (0.00)
  Diarrhoea: Week 96: number analyzed (Participants) | 2
  Diarrhoea: Week 96 | 33.33 (47.14)
  Diarrhoea: Week 99: number analyzed (Participants) | 1
  Diarrhoea: Week 99 | 0.00
  Diarrhoea: Week 105: number analyzed (Participants) | 1
  Diarrhoea: Week 105 | 0.00
  Diarrhoea: Week 111: number analyzed (Participants) | 1
  Diarrhoea: Week 111 | 0.00
  Diarrhoea: Week 117: number analyzed (Participants) | 1
  Diarrhoea: Week 117 | 0.00
  Diarrhoea: Last visit: number analyzed (Participants) | 72
  Diarrhoea: Last visit | -2.31 (28.15)
  Financial difficulties: Baseline | 30.80 (33.24)
  Financial difficulties: Week 6: number analyzed (Participants) | 64
  Financial difficulties: Week 6 | -2.60 (21.66)
  Financial difficulties: Week 9: number analyzed (Participants) | 1
  Financial difficulties: Week 9 | 0.00
  Financial difficulties: Week 12: number analyzed (Participants) | 54
  Financial difficulties: Week 12 | -4.32 (23.39)
  Financial difficulties: Week 15: number analyzed (Participants) | 1
  Financial difficulties: Week 15 | 0.00
  Financial difficulties: Week 18: number analyzed (Participants) | 49
  Financial difficulties: Week 18 | -4.76 (21.52)
  Financial difficulties: Week 21: number analyzed (Participants) | 1
  Financial difficulties: Week 21 | 0.00
  Financial difficulties: Week 24: number analyzed (Participants) | 41
  Financial difficulties: Week 24 | -2.44 (26.24)
  Financial difficulties: Week 27: number analyzed (Participants) | 2
  Financial difficulties: Week 27 | 0.00 (0.00)
  Financial difficulties: Week 30: number analyzed (Participants) | 39
  Financial difficulties: Week 30 | -6.84 (23.17)
  Financial difficulties: Week 33: number analyzed (Participants) | 3
  Financial difficulties: Week 33 | 11.11 (19.25)
  Financial difficulties: Week 36: number analyzed (Participants) | 38
  Financial difficulties: Week 36 | -6.14 (27.79)
  Financial difficulties: Week 39: number analyzed (Participants) | 2
  Financial difficulties: Week 39 | 16.67 (23.57)
  Financial difficulties: Week 42: number analyzed (Participants) | 36
  Financial difficulties: Week 42 | -6.48 (20.81)
  Financial difficulties: Week 45: number analyzed (Participants) | 4
  Financial difficulties: Week 45 | 8.33 (16.67)
  Financial difficulties: Week 48: number analyzed (Participants) | 33
  Financial difficulties: Week 48 | -8.08 (23.61)
  Financial difficulties: Week 51: number analyzed (Participants) | 2
  Financial difficulties: Week 51 | 16.67 (23.57)
  Financial difficulties: Week 54: number analyzed (Participants) | 31
  Financial difficulties: Week 54 | -2.15 (27.13)
  Financial difficulties: Week 57: number analyzed (Participants) | 5
  Financial difficulties: Week 57 | 6.67 (14.91)
  Financial difficulties: Week 60: number analyzed (Participants) | 30
  Financial difficulties: Week 60 | -3.33 (22.06)
  Financial difficulties: Week 63: number analyzed (Participants) | 3
  Financial difficulties: Week 63 | 0.00 (0.00)
  Financial difficulties: Week 66: number analyzed (Participants) | 26
  Financial difficulties: Week 66 | -2.56 (28.16)
  Financial difficulties: Week 69: number analyzed (Participants) | 4
  Financial difficulties: Week 69 | -8.33 (16.67)
  Financial difficulties: Week 72: number analyzed (Participants) | 23
  Financial difficulties: Week 72 | 5.80 (25.92)
  Financial difficulties: Week 75: number analyzed (Participants) | 2
  Financial difficulties: Week 75 | 0.00 (0.00)
  Financial difficulties: Week 78: number analyzed (Participants) | 21
  Financial difficulties: Week 78 | 0.00 (34.96)
  Financial difficulties: Week 81: number analyzed (Participants) | 2
  Financial difficulties: Week 81 | 0.00 (0.00)
  Financial difficulties: Week 84: number analyzed (Participants) | 13
  Financial difficulties: Week 84 | 12.82 (34.80)
  Financial difficulties: Week 87: number analyzed (Participants) | 3
  Financial difficulties: Week 87 | 0.00 (0.00)
  Financial difficulties: Week 90: number analyzed (Participants) | 8
  Financial difficulties: Week 90 | -4.17 (21.36)
  Financial difficulties: Week 93: number analyzed (Participants) | 2
  Financial difficulties: Week 93 | -16.67 (23.57)
  Financial difficulties: Week 96: number analyzed (Participants) | 3
  Financial difficulties: Week 96 | 22.22 (38.49)
  Financial difficulties: Week 99: number analyzed (Participants) | 1
  Financial difficulties: Week 99 | 0.00
  Financial difficulties: Week 105: number analyzed (Participants) | 1
  Financial difficulties: Week 105 | 0.00
  Financial difficulties: Week 111: number analyzed (Participants) | 1
  Financial difficulties: Week 111 | 0.00
  Financial difficulties: Week 117: number analyzed (Participants) | 1
  Financial difficulties: Week 117 | 0.00
  Financial difficulties: Last visit: number analyzed (Participants) | 73
  Financial difficulties: Last visit | 1.83 (32.82)

28. Secondary Outcome: Change From Baseline in EORTC Quality of Life Questionnaire Lung Cancer 13 (EORTC QLQ-LC13): Phase II
Description: EORTC QLQ-LC13 consisted of 13 questions for dyspnea (3 items) and 10 single items (cough, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in chest, pain in arm/shoulder, other pain). Questions used 4-point scale (1 'Not at all' to 4 'Very much'). Scores were averaged and transformed to 0-100 scale; higher score=better level of functioning, lower score indicates lower level of functioning. 'Baseline' category for any parameter below represents absolute data at baseline.
Time Frame: as for outcome 27
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alectinib 600 mg (Fed): Phase II
Number analyzed (Participants) | 79
units on a scale
  Dyspnoea: Baseline: number analyzed (Participants) | 76
  Dyspnoea: Baseline | 30.85 (27.13)
  Dyspnoea: Week 6: number analyzed (Participants) | 58
  Dyspnoea: Week 6 | -8.24 (22.57)
  Dyspnoea: Week 9: number analyzed (Participants) | 1
  Dyspnoea: Week 9 | 0.00
  Dyspnoea: Week 12: number analyzed (Participants) | 48
  Dyspnoea: Week 12 | -7.64 (20.65)
  Dyspnoea: Week 15: number analyzed (Participants) | 1
  Dyspnoea: Week 15 | 0.00
  Dyspnoea: Week 18: number analyzed (Participants) | 47
  Dyspnoea: Week 18 | -11.35 (21.67)
  Dyspnoea: Week 21: number analyzed (Participants) | 1
  Dyspnoea: Week 21 | 0.00
  Dyspnoea: Week 24: number analyzed (Participants) | 39
  Dyspnoea: Week 24 | -7.41 (21.68)
  Dyspnoea: Week 27: number analyzed (Participants) | 2
  Dyspnoea: Week 27 | 5.56 (7.86)
  Dyspnoea: Week 30: number analyzed (Participants) | 38
  Dyspnoea: Week 30 | -4.09 (20.41)
  Dyspnoea: Week 33: number analyzed (Participants) | 3
  Dyspnoea: Week 33 | -11.11 (11.11)
  Dyspnoea: Week 36: number analyzed (Participants) | 37
  Dyspnoea: Week 36 | -5.41 (21.69)
  Dyspnoea: Week 39: number analyzed (Participants) | 2
  Dyspnoea: Week 39 | -5.56 (7.86)
  Dyspnoea: Week 42: number analyzed (Participants) | 36
  Dyspnoea: Week 42 | -8.64 (20.25)
  Dyspnoea: Week 45: number analyzed (Participants) | 4
  Dyspnoea: Week 45 | -2.78 (27.78)
  Dyspnoea: Week 48: number analyzed (Participants) | 33
  Dyspnoea: Week 48 | -7.74 (24.77)
  Dyspnoea: Week 51: number analyzed (Participants) | 2
  Dyspnoea: Week 51 | -27.78 (23.57)
  Dyspnoea: Week 54: number analyzed (Participants) | 31
  Dyspnoea: Week 54 | -5.02 (19.63)
  Dyspnoea: Week 57: number analyzed (Participants) | 5
  Dyspnoea: Week 57 | -2.22 (16.48)
  Dyspnoea: Week 60: number analyzed (Participants) | 29
  Dyspnoea: Week 60 | -7.28 (19.54)
  Dyspnoea: Week 63: number analyzed (Participants) | 3
  Dyspnoea: Week 63 | 3.70 (16.97)
  Dyspnoea: Week 66: number analyzed (Participants) | 25
  Dyspnoea: Week 66 | -6.22 (25.27)
  Dyspnoea: Week 69: number analyzed (Participants) | 4
  Dyspnoea: Week 69 | -13.89 (29.22)
  Dyspnoea: Week 72: number analyzed (Participants) | 23
  Dyspnoea: Week 72 | -6.76 (26.96)
  Dyspnoea: Week 75: number analyzed (Participants) | 2
  Dyspnoea: Week 75 | -5.56 (7.86)
  Dyspnoea: Week 78: number analyzed (Participants) | 19
  Dyspnoea: Week 78 | -8.19 (22.48)
  Dyspnoea: Week 81: number analyzed (Participants) | 2
  Dyspnoea: Week 81 | -5.56 (7.86)
  Dyspnoea: Week 84: number analyzed (Participants) | 13
  Dyspnoea: Week 84 | -9.40 (16.26)
  Dyspnoea: Week 87: number analyzed (Participants) | 3
  Dyspnoea: Week 87 | 7.41 (23.13)
  Dyspnoea: Week 90: number analyzed (Participants) | 8
  Dyspnoea: Week 90 | -5.56 (17.82)
  Dyspnoea: Week 93: number analyzed (Participants) | 2
  Dyspnoea: Week 93 | 22.22 (0.00)
  Dyspnoea: Week 96: number analyzed (Participants) | 3
  Dyspnoea: Week 96 | -51.85 (23.13)
  Dyspnoea: Week 99: number analyzed (Participants) | 1
  Dyspnoea: Week 99 | 11.11
  Dyspnoea: Week 105: number analyzed (Participants) | 1
  Dyspnoea: Week 105 | 0.00
  Dyspnoea: Week 111: number analyzed (Participants) | 1
  Dyspnoea: Week 111 | 0.00
  Dyspnoea: Week 117: number analyzed (Participants) | 1
  Dyspnoea: Week 117 | 0.00
  Dyspnoea: Last visit: number analyzed (Participants) | 69
  Dyspnoea: Last visit | -6.44 (23.45)
  Coughing: Baseline | 33.76 (27.47)
  Coughing: Week 6: number analyzed (Participants) | 60
  Coughing: Week 6 | -13.89 (31.47)
  Coughing: Week 9: number analyzed (Participants) | 1
  Coughing: Week 9 | 0.00
  Coughing: Week 12: number analyzed (Participants) | 52
  Coughing: Week 12 | -12.82 (27.34)
  Coughing: Week 15: number analyzed (Participants) | 1
  Coughing: Week 15 | 0.00
  Coughing: Week 18: number analyzed (Participants) | 49
  Coughing: Week 18 | -13.61 (24.46)
  Coughing: Week 21: number analyzed (Participants) | 1
  Coughing: Week 21 | 0.00
  Coughing: Week 24: number analyzed (Participants) | 40
  Coughing: Week 24 | -9.17 (31.11)
  Coughing: Week 27: number analyzed (Participants) | 2
  Coughing: Week 27 | 0.00 (0.00)
  Coughing: Week 30: number analyzed (Participants) | 38
  Coughing: Week 30 | -1.75 (24.44)
  Coughing: Week 33: number analyzed (Participants) | 3
  Coughing: Week 33 | -22.22 (19.25)
  Coughing: Week 36: number analyzed (Participants) | 38
  Coughing: Week 36 | -8.77 (28.67)
  Coughing: Week 39: number analyzed (Participants) | 2
  Coughing: Week 39 | -50.00 (23.57)
  Coughing: Week 42: number analyzed (Participants) | 36
  Coughing: Week 42 | -0.93 (27.01)
  Coughing: Week 45: number analyzed (Participants) | 4
  Coughing: Week 45 | -8.33 (50.00)
  Coughing: Week 48: number analyzed (Participants) | 33
  Coughing: Week 48 | -4.04 (35.12)
  Coughing: Week 51: number analyzed (Participants) | 2
  Coughing: Week 51 | -33.33 (0.00)
  Coughing: Week 54: number analyzed (Participants) | 32
  Coughing: Week 54 | -8.33 (25.40)
  Coughing: Week 57: number analyzed (Participants) | 5
  Coughing: Week 57 | -20.00 (29.81)
  Coughing: Week 60: number analyzed (Participants) | 29
  Coughing: Week 60 | -2.30 (29.45)
  Coughing: Week 63: number analyzed (Participants) | 3
  Coughing: Week 63 | 0.00 (33.33)
  Coughing: Week 66: number analyzed (Participants) | 26
  Coughing: Week 66 | -5.13 (27.80)
  Coughing: Week 69: number analyzed (Participants) | 4
  Coughing: Week 69 | -25.00 (31.91)
  Coughing: Week 72: number analyzed (Participants) | 23
  Coughing: Week 72 | -7.25 (28.35)
  Coughing: Week 75: number analyzed (Participants) | 2
  Coughing: Week 75 | -16.67 (23.57)
  Coughing: Week 78: number analyzed (Participants) | 20
  Coughing: Week 78 | -6.67 (35.21)
  Coughing: Week 81: number analyzed (Participants) | 2
  Coughing: Week 81 | -16.67 (23.57)
  Coughing: Week 84: number analyzed (Participants) | 13
  Coughing: Week 84 | -15.38 (29.24)
  Coughing: Week 87: number analyzed (Participants) | 3
  Coughing: Week 87 | 0.00 (33.33)
  Coughing: Week 90: number analyzed (Participants) | 8
  Coughing: Week 90 | -8.33 (29.55)
  Coughing: Week 93: number analyzed (Participants) | 2
  Coughing: Week 93 | 16.67 (23.57)
  Coughing: Week 96: number analyzed (Participants) | 3
  Coughing: Week 96 | -44.44 (19.25)
  Coughing: Week 99: number analyzed (Participants) | 1
  Coughing: Week 99 | 0.00
  Coughing: Week 105: number analyzed (Participants) | 1
  Coughing: Week 105 | 0.00
  Coughing: Week 111: number analyzed (Participants) | 1
  Coughing: Week 111 | 0.00
  Coughing: Week 117: number analyzed (Participants) | 1
  Coughing: Week 117 | 0.00
  Coughing: Last visit: number analyzed (Participants) | 73
  Coughing: Last visit | -5.48 (32.87)
  Hemoptysis: Baseline | 1.27 (6.41)
  Hemoptysis: Week 6: number analyzed (Participants) | 60
  Hemoptysis: Week 6 | -1.11 (6.03)
  Hemoptysis: Week 9: number analyzed (Participants) | 1
  Hemoptysis: Week 9 | 0.00
  Hemoptysis: Week 12: number analyzed (Participants) | 52
  Hemoptysis: Week 12 | -1.28 (6.47)
  Hemoptysis: Week 15: number analyzed (Participants) | 1
  Hemoptysis: Week 15 | 0.00
  Hemoptysis: Week 18: number analyzed (Participants) | 49
  Hemoptysis: Week 18 | -1.36 (6.66)
  Hemoptysis: Week 21: number analyzed (Participants) | 1
  Hemoptysis: Week 21 | 0.00
  Hemoptysis: Week 24: number analyzed (Participants) | 40
  Hemoptysis: Week 24 | -1.67 (7.36)
  Hemoptysis: Week 27: number analyzed (Participants) | 2
  Hemoptysis: Week 27 | 0.00 (0.00)
  Hemoptysis: Week 30: number analyzed (Participants) | 39
  Hemoptysis: Week 30 | 0.00 (13.25)
  Hemoptysis: Week 33: number analyzed (Participants) | 3
  Hemoptysis: Week 33 | 0.00 (0.00)
  Hemoptysis: Week 36: number analyzed (Participants) | 38
  Hemoptysis: Week 36 | -1.75 (7.54)
  Hemoptysis: Week 39: number analyzed (Participants) | 2
  Hemoptysis: Week 39 | 0.00 (0.00)
  Hemoptysis: Week 42: number analyzed (Participants) | 36
  Hemoptysis: Week 42 | 0.00 (7.97)
  Hemoptysis: Week 45: number analyzed (Participants) | 4
  Hemoptysis: Week 45 | 0.00 (0.00)
  Hemoptysis: Week 48: number analyzed (Participants) | 33
  Hemoptysis: Week 48 | -1.01 (5.80)
  Hemoptysis: Week 51: number analyzed (Participants) | 2
  Hemoptysis: Week 51 | 0.00 (0.00)
  Hemoptysis: Week 54: number analyzed (Participants) | 31
  Hemoptysis: Week 54 | 1.08 (10.48)
  Hemoptysis: Week 57: number analyzed (Participants) | 5
  Hemoptysis: Week 57 | 0.00 (0.00)
  Hemoptysis: Week 60: number analyzed (Participants) | 29
  Hemoptysis: Week 60 | -1.15 (6.19)
  Hemoptysis: Week 63: number analyzed (Participants) | 3
  Hemoptysis: Week 63 | 0.00 (0.00)
  Hemoptysis: Week 66: number analyzed (Participants) | 26
  Hemoptysis: Week 66 | -1.28 (6.54)
  Hemoptysis: Week 69: number analyzed (Participants) | 4
  Hemoptysis: Week 69 | 0.00 (0.00)
  Hemoptysis: Week 72: number analyzed (Participants) | 23
  Hemoptysis: Week 72 | 2.90 (22.28)
  Hemoptysis: Week 75: number analyzed (Participants) | 2
  Hemoptysis: Week 75 | 0.00 (0.00)
  Hemoptysis: Week 78: number analyzed (Participants) | 20
  Hemoptysis: Week 78 | -1.67 (7.45)
  Hemoptysis: Week 81: number analyzed (Participants) | 2
  Hemoptysis: Week 81 | 0.00 (0.00)
  Hemoptysis: Week 84: number analyzed (Participants) | 13
  Hemoptysis: Week 84 | -2.56 (9.25)
  Hemoptysis: Week 87: number analyzed (Participants) | 3
  Hemoptysis: Week 87 | 0.00 (0.00)
  Hemoptysis: Week 90: number analyzed (Participants) | 8
  Hemoptysis: Week 90 | 0.00 (0.00)
  Hemoptysis: Week 93: number analyzed (Participants) | 2
  Hemoptysis: Week 93 | 0.00 (0.00)
  Hemoptysis: Week 96: number analyzed (Participants) | 3
  Hemoptysis: Week 96 | 0.00 (0.00)
  Hemoptysis: Week 99: number analyzed (Participants) | 1
  Hemoptysis: Week 99 | 0.00
  Hemoptysis: Week 105: number analyzed (Participants) | 1
  Hemoptysis: Week 105 | 0.00
  Hemoptysis: Week 111: number analyzed (Participants) | 1
  Hemoptysis: Week 111 | 0.00
  Hemoptysis: Week 117: number analyzed (Participants) | 1
  Hemoptysis: Week 117 | 0.00
  Hemoptysis: Last visit: number analyzed (Participants) | 73
  Hemoptysis: Last visit | -0.91 (7.80)
  Sore mouth: Baseline | 5.06 (16.09)
  Sore mouth: Week 6: number analyzed (Participants) | 60
  Sore mouth: Week 6 | -1.11 (13.68)
  Sore mouth: Week 9: number analyzed (Participants) | 1
  Sore mouth: Week 9 | 0.00
  Sore mouth: Week 12: number analyzed (Participants) | 52
  Sore mouth: Week 12 | 0.64 (13.99)
  Sore mouth: Week 15: number analyzed (Participants) | 1
  Sore mouth: Week 15 | 0.00
  Sore mouth: Week 18: number analyzed (Participants) | 49
  Sore mouth: Week 18 | -2.04 (17.22)
  Sore mouth: Week 21: number analyzed (Participants) | 1
  Sore mouth: Week 21 | 0.00
  Sore mouth: Week 24: number analyzed (Participants) | 39
  Sore mouth: Week 24 | -0.85 (17.91)
  Sore mouth: Week 27: number analyzed (Participants) | 2
  Sore mouth: Week 27 | 0.00 (0.00)
  Sore mouth: Week 30: number analyzed (Participants) | 39
  Sore mouth: Week 30 | 2.56 (11.81)
  Sore mouth: Week 33: number analyzed (Participants) | 3
  Sore mouth: Week 33 | 22.22 (38.49)
  Sore mouth: Week 36: number analyzed (Participants) | 38
  Sore mouth: Week 36 | 1.75 (15.40)
  Sore mouth: Week 39: number analyzed (Participants) | 2
  Sore mouth: Week 39 | 16.67 (23.57)
  Sore mouth: Week 42: number analyzed (Participants) | 36
  Sore mouth: Week 42 | -0.93 (9.71)
  Sore mouth: Week 45: number analyzed (Participants) | 4
  Sore mouth: Week 45 | 0.00 (0.00)
  Sore mouth: Week 48: number analyzed (Participants) | 33
  Sore mouth: Week 48 | 7.07 (26.03)
  Sore mouth: Week 51: number analyzed (Participants) | 2
  Sore mouth: Week 51 | 0.00 (0.00)
  Sore mouth: Week 54: number analyzed (Participants) | 31
  Sore mouth: Week 54 | 1.08 (13.56)
  Sore mouth: Week 57: number analyzed (Participants) | 5
  Sore mouth: Week 57 | 0.00 (23.57)
  Sore mouth: Week 60: number analyzed (Participants) | 29
  Sore mouth: Week 60 | -1.15 (14.04)
  Sore mouth: Week 63: number analyzed (Participants) | 3
  Sore mouth: Week 63 | 0.00 (0.00)
  Sore mouth: Week 66: number analyzed (Participants) | 26
  Sore mouth: Week 66 | -2.56 (13.07)
  Sore mouth: Week 69: number analyzed (Participants) | 4
  Sore mouth: Week 69 | 0.00 (0.00)
  Sore mouth: Week 72: number analyzed (Participants) | 22
  Sore mouth: Week 72 | 4.55 (18.67)
  Sore mouth: Week 75: number analyzed (Participants) | 2
  Sore mouth: Week 75 | 0.00 (0.00)
  Sore mouth: Week 78: number analyzed (Participants) | 20
  Sore mouth: Week 78 | 1.67 (7.45)
  Sore mouth: Week 81: number analyzed (Participants) | 2
  Sore mouth: Week 81 | 0.00 (0.00)
  Sore mouth: Week 84: number analyzed (Participants) | 13
  Sore mouth: Week 84 | 0.00 (0.00)
  Sore mouth: Week 87: number analyzed (Participants) | 3
  Sore mouth: Week 87 | 0.00 (0.00)
  Sore mouth: Week 90: number analyzed (Participants) | 8
  Sore mouth: Week 90 | 4.17 (11.79)
  Sore mouth: Week 93: number analyzed (Participants) | 2
  Sore mouth: Week 93 | 0.00 (0.00)
  Sore mouth: Week 96: number analyzed (Participants) | 3
  Sore mouth: Week 96 | 11.11 (19.25)
  Sore mouth: Week 99: number analyzed (Participants) | 1
  Sore mouth: Week 99 | 0.00
  Sore mouth: Week 105: number analyzed (Participants) | 1
  Sore mouth: Week 105 | 0.00
  Sore mouth: Week 111: number analyzed (Participants) | 1
  Sore mouth: Week 111 | 0.00
  Sore mouth: Week 117: number analyzed (Participants) | 1
  Sore mouth: Week 117 | 0.00
  Sore mouth: Last visit: number analyzed (Participants) | 73
  Sore mouth: Last visit | -0.46 (15.21)
  Dysphagia: Baseline | 4.64 (11.61)
  Dysphagia: Week 6: number analyzed (Participants) | 60
  Dysphagia: Week 6 | -1.67 (11.36)
  Dysphagia: Week 9: number analyzed (Participants) | 1
  Dysphagia: Week 9 | 0.00
  Dysphagia: Week 12: number analyzed (Participants) | 52
  Dysphagia: Week 12 | -0.64 (10.42)
  Dysphagia: Week 15: number analyzed (Participants) | 1
  Dysphagia: Week 15 | 0.00
  Dysphagia: Week 18: number analyzed (Participants) | 49
  Dysphagia: Week 18 | -1.36 (11.70)
  Dysphagia: Week 21: number analyzed (Participants) | 1
  Dysphagia: Week 21 | 0.00
  Dysphagia: Week 24: number analyzed (Participants) | 40
  Dysphagia: Week 24 | 0.83 (11.91)
  Dysphagia: Week 27: number analyzed (Participants) | 2
  Dysphagia: Week 27 | 16.67 (23.57)
  Dysphagia: Week 30: number analyzed (Participants) | 39
  Dysphagia: Week 30 | 3.42 (14.90)
  Dysphagia: Week 33: number analyzed (Participants) | 3
  Dysphagia: Week 33 | 0.00 (33.33)
  Dysphagia: Week 36: number analyzed (Participants) | 38
  Dysphagia: Week 36 | -0.88 (5.41)
  Dysphagia: Week 39: number analyzed (Participants) | 2
  Dysphagia: Week 39 | -16.67 (23.57)
  Dysphagia: Week 42: number analyzed (Participants) | 36
  Dysphagia: Week 42 | -0.93 (12.56)
  Dysphagia: Week 45: number analyzed (Participants) | 4
  Dysphagia: Week 45 | 0.00 (27.22)
  Dysphagia: Week 48: number analyzed (Participants) | 33
  Dysphagia: Week 48 | 2.02 (16.54)
  Dysphagia: Week 51: number analyzed (Participants) | 2
  Dysphagia: Week 51 | -16.67 (23.57)
  Dysphagia: Week 54: number analyzed (Participants) | 31
  Dysphagia: Week 54 | -1.08 (13.56)
  Dysphagia: Week 57: number analyzed (Participants) | 5
  Dysphagia: Week 57 | 6.67 (27.89)
  Dysphagia: Week 60: number analyzed (Participants) | 28
  Dysphagia: Week 60 | -3.57 (13.88)
  Dysphagia: Week 63: number analyzed (Participants) | 3
  Dysphagia: Week 63 | 11.11 (19.25)
  Dysphagia: Week 66: number analyzed (Participants) | 26
  Dysphagia: Week 66 | -1.28 (14.85)
  Dysphagia: Week 69: number analyzed (Participants) | 4
  Dysphagia: Week 69 | 0.00 (0.00)
  Dysphagia: Week 72: number analyzed (Participants) | 23
  Dysphagia: Week 72 | 1.45 (15.82)
  Dysphagia: Week 75: number analyzed (Participants) | 2
  Dysphagia: Week 75 | 0.00 (0.00)
  Dysphagia: Week 78: number analyzed (Participants) | 20
  Dysphagia: Week 78 | 0.00 (10.81)
  Dysphagia: Week 81: number analyzed (Participants) | 2
  Dysphagia: Week 81 | 0.00 (0.00)
  Dysphagia: Week 84: number analyzed (Participants) | 13
  Dysphagia: Week 84 | 2.56 (9.25)
  Dysphagia: Week 87: number analyzed (Participants) | 3
  Dysphagia: Week 87 | 0.00 (0.00)
  Dysphagia: Week 90: number analyzed (Participants) | 8
  Dysphagia: Week 90 | 0.00 (0.00)
  Dysphagia: Week 93: number analyzed (Participants) | 2
  Dysphagia: Week 93 | 0.00 (0.00)
  Dysphagia: Week 96: number analyzed (Participants) | 3
  Dysphagia: Week 96 | 0.00 (0.00)
  Dysphagia: Week 99: number analyzed (Participants) | 1
  Dysphagia: Week 99 | 0.00
  Dysphagia: Week 105: number analyzed (Participants) | 1
  Dysphagia: Week 105 | 0.00
  Dysphagia: Week 111: number analyzed (Participants) | 1
  Dysphagia: Week 111 | 0.00
  Dysphagia: Week 117: number analyzed (Participants) | 1
  Dysphagia: Week 117 | 0.00
  Dysphagia: Last visit: number analyzed (Participants) | 73
  Dysphagia: Last visit | 2.74 (17.35)
  Peripheral neuropathy: Baseline | 13.08 (22.28)
  Peripheral neuropathy: Week 6: number analyzed (Participants) | 60
  Peripheral neuropathy: Week 6 | 6.11 (17.88)
  Peripheral neuropathy: Week 9: number analyzed (Participants) | 1
  Peripheral neuropathy: Week 9 | 0.00
  Peripheral neuropathy: Week 12: number analyzed (Participants) | 52
  Peripheral neuropathy: Week 12 | 1.28 (20.83)
  Peripheral neuropathy: Week 15: number analyzed (Participants) | 1
  Peripheral neuropathy: Week 15 | 0.00
  Peripheral neuropathy: Week 18: number analyzed (Participants) | 49
  Peripheral neuropathy: Week 18 | 2.72 (22.40)
  Peripheral neuropathy: Week 21: number analyzed (Participants) | 1
  Peripheral neuropathy: Week 21 | 0.00
  Peripheral neuropathy: Week 24: number analyzed (Participants) | 40
  Peripheral neuropathy: Week 24 | 4.17 (20.24)
  Peripheral neuropathy: Week 27: number analyzed (Participants) | 2
  Peripheral neuropathy: Week 27 | -16.67 (23.57)
  Peripheral neuropathy: Week 30: number analyzed (Participants) | 39
  Peripheral neuropathy: Week 30 | 4.27 (24.40)
  Peripheral neuropathy: Week 33: number analyzed (Participants) | 3
  Peripheral neuropathy: Week 33 | 11.11 (19.25)
  Peripheral neuropathy: Week 36: number analyzed (Participants) | 38
  Peripheral neuropathy: Week 36 | 0.00 (18.98)
  Peripheral neuropathy: Week 39: number analyzed (Participants) | 2
  Peripheral neuropathy: Week 39 | 0.00 (0.00)
  Peripheral neuropathy: Week 42: number analyzed (Participants) | 36
  Peripheral neuropathy: Week 42 | 1.85 (21.00)
  Peripheral neuropathy: Week 45: number analyzed (Participants) | 4
  Peripheral neuropathy: Week 45 | 8.33 (16.67)
  Peripheral neuropathy: Week 48: number analyzed (Participants) | 33
  Peripheral neuropathy: Week 48 | 2.02 (23.48)
  Peripheral neuropathy: Week 51: number analyzed (Participants) | 2
  Peripheral neuropathy: Week 51 | 0.00 (0.00)
  Peripheral neuropathy: Week 54: number analyzed (Participants) | 31
  Peripheral neuropathy: Week 54 | 6.45 (26.41)
  Peripheral neuropathy: Week 57: number analyzed (Participants) | 5
  Peripheral neuropathy: Week 57 | 6.67 (27.89)
  Peripheral neuropathy: Week 60: number analyzed (Participants) | 29
  Peripheral neuropathy: Week 60 | 2.30 (23.45)
  Peripheral neuropathy: Week 63: number analyzed (Participants) | 3
  Peripheral neuropathy: Week 63 | 0.00 (0.00)
  Peripheral neuropathy: Week 66: number analyzed (Participants) | 26
  Peripheral neuropathy: Week 66 | 1.28 (24.00)
  Peripheral neuropathy: Week 69: number analyzed (Participants) | 4
  Peripheral neuropathy: Week 69 | 0.00 (0.00)
  Peripheral neuropathy: Week 72: number analyzed (Participants) | 23
  Peripheral neuropathy: Week 72 | 2.90 (28.27)
  Peripheral neuropathy: Week 75: number analyzed (Participants) | 2
  Peripheral neuropathy: Week 75 | 0.00 (0.00)
  Peripheral neuropathy: Week 78: number analyzed (Participants) | 20
  Peripheral neuropathy: Week 78 | -3.33 (21.36)
  Peripheral neuropathy: Week 81: number analyzed (Participants) | 2
  Peripheral neuropathy: Week 81 | 0.00 (0.00)
  Peripheral neuropathy: Week 84: number analyzed (Participants) | 13
  Peripheral neuropathy: Week 84 | 12.82 (37.36)
  Peripheral neuropathy: Week 87: number analyzed (Participants) | 3
  Peripheral neuropathy: Week 87 | 0.00 (0.00)
  Peripheral neuropathy: Week 90: number analyzed (Participants) | 8
  Peripheral neuropathy: Week 90 | 16.67 (17.82)
  Peripheral neuropathy: Week 93: number analyzed (Participants) | 2
  Peripheral neuropathy: Week 93 | 0.00 (0.00)
  Peripheral neuropathy: Week 96: number analyzed (Participants) | 3
  Peripheral neuropathy: Week 96 | 55.56 (38.49)
  Peripheral neuropathy: Week 99: number analyzed (Participants) | 1
  Peripheral neuropathy: Week 99 | 0.00
  Peripheral neuropathy: Week 105: number analyzed (Participants) | 1
  Peripheral neuropathy: Week 105 | 0.00
  Peripheral neuropathy: Week 111: number analyzed (Participants) | 1
  Peripheral neuropathy: Week 111 | 0.00
  Peripheral neuropathy: Week 117: number analyzed (Participants) | 1
  Peripheral neuropathy: Week 117 | 0.00
  Peripheral neuropathy: Last visit: number analyzed (Participants) | 73
  Peripheral neuropathy: Last visit | 1.37 (22.52)
  Alopecia: Baseline: number analyzed (Participants) | 77
  Alopecia: Baseline | 11.69 (25.80)
  Alopecia: Week 6: number analyzed (Participants) | 59
  Alopecia: Week 6 | -1.13 (22.29)
  Alopecia: Week 9: number analyzed (Participants) | 1
  Alopecia: Week 9 | 0.00
  Alopecia: Week 12: number analyzed (Participants) | 51
  Alopecia: Week 12 | 1.31 (31.24)
  Alopecia: Week 15: number analyzed (Participants) | 1
  Alopecia: Week 15 | 0.00
  Alopecia: Week 18: number analyzed (Participants) | 47
  Alopecia: Week 18 | -4.96 (25.04)
  Alopecia: Week 21: number analyzed (Participants) | 1
  Alopecia: Week 21 | 0.00
  Alopecia: Week 24: number analyzed (Participants) | 39
  Alopecia: Week 24 | -2.56 (27.98)
  Alopecia: Week 27: number analyzed (Participants) | 2
  Alopecia: Week 27 | 0.00 (0.00)
  Alopecia: Week 30: number analyzed (Participants) | 38
  Alopecia: Week 30 | -3.51 (27.72)
  Alopecia: Week 33: number analyzed (Participants) | 3
  Alopecia: Week 33 | 0.00 (0.00)
  Alopecia: Week 36: number analyzed (Participants) | 37
  Alopecia: Week 36 | 0.90 (32.85)
  Alopecia: Week 39: number analyzed (Participants) | 2
  Alopecia: Week 39 | 0.00 (0.00)
  Alopecia: Week 42: number analyzed (Participants) | 36
  Alopecia: Week 42 | -2.78 (20.12)
  Alopecia: Week 45: number analyzed (Participants) | 4
  Alopecia: Week 45 | 0.00 (0.00)
  Alopecia: Week 48: number analyzed (Participants) | 32
  Alopecia: Week 48 | -5.21 (22.58)
  Alopecia: Week 51: number analyzed (Participants) | 2
  Alopecia: Week 51 | 0.00 (0.00)
  Alopecia: Week 54: number analyzed (Participants) | 31
  Alopecia: Week 54 | -6.45 (15.91)
  Alopecia: Week 57: number analyzed (Participants) | 5
  Alopecia: Week 57 | -6.67 (14.91)
  Alopecia: Week 60: number analyzed (Participants) | 29
  Alopecia: Week 60 | -4.60 (19.36)
  Alopecia: Week 63: number analyzed (Participants) | 3
  Alopecia: Week 63 | -11.11 (19.25)
  Alopecia: Week 66: number analyzed (Participants) | 25
  Alopecia: Week 66 | -2.67 (27.08)
  Alopecia: Week 69: number analyzed (Participants) | 4
  Alopecia: Week 69 | -8.33 (16.67)
  Alopecia: Week 72: number analyzed (Participants) | 22
  Alopecia: Week 72 | -3.03 (33.98)
  Alopecia: Week 75: number analyzed (Participants) | 2
  Alopecia: Week 75 | 0.00 (0.00)
  Alopecia: Week 78: number analyzed (Participants) | 20
  Alopecia: Week 78 | -8.33 (26.21)
  Alopecia: Week 81: number analyzed (Participants) | 2
  Alopecia: Week 81 | -16.67 (23.57)
  Alopecia: Week 84: number analyzed (Participants) | 13
  Alopecia: Week 84 | -2.56 (25.32)
  Alopecia: Week 87: number analyzed (Participants) | 3
  Alopecia: Week 87 | -11.11 (19.25)
  Alopecia: Week 90: number analyzed (Participants) | 8
  Alopecia: Week 90 | 4.17 (21.36)
  Alopecia: Week 93: number analyzed (Participants) | 2
  Alopecia: Week 93 | 0.00 (0.00)
  Alopecia: Week 96: number analyzed (Participants) | 3
  Alopecia: Week 96 | 0.00 (0.00)
  Alopecia: Week 99: number analyzed (Participants) | 1
  Alopecia: Week 99 | 0.00
  Alopecia: Week 105: number analyzed (Participants) | 1
  Alopecia: Week 105 | 0.00
  Alopecia: Week 111: number analyzed (Participants) | 1
  Alopecia: Week 111 | 0.00
  Alopecia: Week 117: number analyzed (Participants) | 1
  Alopecia: Week 117 | 0.00
  Alopecia: Last visit: number analyzed (Participants) | 71
  Alopecia: Last visit | -5.16 (27.97)
  Pain in chest: Baseline | 21.52 (28.26)
  Pain in chest: Week 6: number analyzed (Participants) | 60
  Pain in chest: Week 6 | -16.67 (29.75)
  Pain in chest: Week 9: number analyzed (Participants) | 1
  Pain in chest: Week 9 | 0.00
  Pain in chest: Week 12: number analyzed (Participants) | 52
  Pain in chest: Week 12 | -11.54 (23.69)
  Pain in chest: Week 15: number analyzed (Participants) | 1
  Pain in chest: Week 15 | 0.00
  Pain in chest: Week 18: number analyzed (Participants) | 49
  Pain in chest: Week 18 | -8.84 (27.87)
  Pain in chest: Week 21: number analyzed (Participants) | 1
  Pain in chest: Week 21 | 0.00
  Pain in chest: Week 24: number analyzed (Participants) | 40
  Pain in chest: Week 24 | -8.33 (23.57)
  Pain in chest: Week 27: number analyzed (Participants) | 2
  Pain in chest: Week 27 | 0.00 (0.00)
  Pain in chest: Week 30: number analyzed (Participants) | 39
  Pain in chest: Week 30 | -3.42 (22.68)
  Pain in chest: Week 33: number analyzed (Participants) | 3
  Pain in chest: Week 33 | -11.11 (19.25)
  Pain in chest: Week 36: number analyzed (Participants) | 38
  Pain in chest: Week 36 | -6.14 (26.68)
  Pain in chest: Week 39: number analyzed (Participants) | 2
  Pain in chest: Week 39 | -16.67 (23.57)
  Pain in chest: Week 42: number analyzed (Participants) | 36
  Pain in chest: Week 42 | -6.48 (19.22)
  Pain in chest: Week 45: number analyzed (Participants) | 4
  Pain in chest: Week 45 | -8.33 (41.94)
  Pain in chest: Week 48: number analyzed (Participants) | 33
  Pain in chest: Week 48 | -6.06 (19.46)
  Pain in chest: Week 51: number analyzed (Participants) | 2
  Pain in chest: Week 51 | -33.33 (0.00)
  Pain in chest: Week 54: number analyzed (Participants) | 31
  Pain in chest: Week 54 | -4.30 (20.62)
  Pain in chest: Week 57: number analyzed (Participants) | 5
  Pain in chest: Week 57 | -13.33 (38.01)
  Pain in chest: Week 60: number analyzed (Participants) | 29
  Pain in chest: Week 60 | -3.45 (16.29)
  Pain in chest: Week 63: number analyzed (Participants) | 2
  Pain in chest: Week 63 | -16.67 (23.57)
  Pain in chest: Week 66: number analyzed (Participants) | 26
  Pain in chest: Week 66 | -2.56 (18.67)
  Pain in chest: Week 69: number analyzed (Participants) | 4
  Pain in chest: Week 69 | -25.00 (31.91)
  Pain in chest: Week 72: number analyzed (Participants) | 23
  Pain in chest: Week 72 | -2.90 (28.27)
  Pain in chest: Week 75: number analyzed (Participants) | 2
  Pain in chest: Week 75 | -16.67 (23.57)
  Pain in chest: Week 78: number analyzed (Participants) | 20
  Pain in chest: Week 78 | 0.00 (18.73)
  Pain in chest: Week 81: number analyzed (Participants) | 2
  Pain in chest: Week 81 | -16.67 (23.57)
  Pain in chest: Week 84: number analyzed (Participants) | 13
  Pain in chest: Week 84 | -5.13 (22.96)
  Pain in chest: Week 87: number analyzed (Participants) | 3
  Pain in chest: Week 87 | -11.11 (19.25)
  Pain in chest: Week 90: number analyzed (Participants) | 8
  Pain in chest: Week 90 | -12.50 (24.80)
  Pain in chest: Week 93: number analyzed (Participants) | 2
  Pain in chest: Week 93 | 16.67 (23.57)
  Pain in chest: Week 96: number analyzed (Participants) | 3
  Pain in chest: Week 96 | -22.22 (19.25)
  Pain in chest: Week 99: number analyzed (Participants) | 1
  Pain in chest: Week 99 | 0.00
  Pain in chest: Week 105: number analyzed (Participants) | 1
  Pain in chest: Week 105 | 0.00
  Pain in chest: Week 111: number analyzed (Participants) | 1
  Pain in chest: Week 111 | 0.00
  Pain in chest: Week 117: number analyzed (Participants) | 1
  Pain in chest: Week 117 | 0.00
  Pain in chest: Last visit: number analyzed (Participants) | 72
  Pain in chest: Last visit | -8.80 (26.83)
  Pain in arm or shoulder: Baseline | 16.88 (28.18)
  Pain in arm or shoulder: Week 6: number analyzed (Participants) | 60
  Pain in arm or shoulder: Week 6 | -7.22 (25.37)
  Pain in arm or shoulder: Week 9: number analyzed (Participants) | 1
  Pain in arm or shoulder: Week 9 | 0.00
  Pain in arm or shoulder: Week 12: number analyzed (Participants) | 52
  Pain in arm or shoulder: Week 12 | -5.77 (30.05)
  Pain in arm or shoulder: Week 15: number analyzed (Participants) | 1
  Pain in arm or shoulder: Week 15 | 0.00
  Pain in arm or shoulder: Week 18: number analyzed (Participants) | 48
  Pain in arm or shoulder: Week 18 | -4.86 (24.78)
  Pain in arm or shoulder: Week 21: number analyzed (Participants) | 1
  Pain in arm or shoulder: Week 21 | 0.00
  Pain in arm or shoulder: Week 24: number analyzed (Participants) | 40
  Pain in arm or shoulder: Week 24 | -10.83 (27.62)
  Pain in arm or shoulder: Week 27: number analyzed (Participants) | 2
  Pain in arm or shoulder: Week 27 | -16.67 (23.57)
  Pain in arm or shoulder: Week 30: number analyzed (Participants) | 39
  Pain in arm or shoulder: Week 30 | -3.42 (23.93)
  Pain in arm or shoulder: Week 33: number analyzed (Participants) | 3
  Pain in arm or shoulder: Week 33 | -11.11 (38.49)
  Pain in arm or shoulder: Week 36: number analyzed (Participants) | 38
  Pain in arm or shoulder: Week 36 | -5.26 (33.36)
  Pain in arm or shoulder: Week 39: number analyzed (Participants) | 2
  Pain in arm or shoulder: Week 39 | -16.67 (23.57)
  Pain in arm or shoulder: Week 42: number analyzed (Participants) | 36
  Pain in arm or shoulder: Week 42 | -5.56 (25.82)
  Pain in arm or shoulder: Week 45: number analyzed (Participants) | 4
  Pain in arm or shoulder: Week 45 | 0.00 (0.00)
  Pain in arm or shoulder: Week 48: number analyzed (Participants) | 33
  Pain in arm or shoulder: Week 48 | -6.06 (21.17)
  Pain in arm or shoulder: Week 51: number analyzed (Participants) | 2
  Pain in arm or shoulder: Week 51 | -16.67 (23.57)
  Pain in arm or shoulder: Week 54: number analyzed (Participants) | 31
  Pain in arm or shoulder: Week 54 | -1.08 (25.07)
  Pain in arm or shoulder: Week 57: number analyzed (Participants) | 5
  Pain in arm or shoulder: Week 57 | 0.00 (23.57)
  Pain in arm or shoulder: Week 60: number analyzed (Participants) | 29
  Pain in arm or shoulder: Week 60 | -2.30 (26.62)
  Pain in arm or shoulder: Week 63: number analyzed (Participants) | 3
  Pain in arm or shoulder: Week 63 | 0.00 (0.00)
  Pain in arm or shoulder: Week 66: number analyzed (Participants) | 26
  Pain in arm or shoulder: Week 66 | -3.85 (27.21)
  Pain in arm or shoulder: Week 69: number analyzed (Participants) | 4
  Pain in arm or shoulder: Week 69 | -16.67 (33.33)
  Pain in arm or shoulder: Week 72: number analyzed (Participants) | 23
  Pain in arm or shoulder: Week 72 | -4.35 (28.96)
  Pain in arm or shoulder: Week 75: number analyzed (Participants) | 2
  Pain in arm or shoulder: Week 75 | 0.00 (0.00)
  Pain in arm or shoulder: Week 78: number analyzed (Participants) | 19
  Pain in arm or shoulder: Week 78 | -8.77 (24.45)
  Pain in arm or shoulder: Week 81: number analyzed (Participants) | 2
  Pain in arm or shoulder: Week 81 | 0.00 (0.00)
  Pain in arm or shoulder: Week 84: number analyzed (Participants) | 13
  Pain in arm or shoulder: Week 84 | 7.69 (38.86)
  Pain in arm or shoulder: Week 87: number analyzed (Participants) | 3
  Pain in arm or shoulder: Week 87 | 0.00 (0.00)
  Pain in arm or shoulder: Week 90: number analyzed (Participants) | 8
  Pain in arm or shoulder: Week 90 | 4.17 (21.36)
  Pain in arm or shoulder: Week 93: number analyzed (Participants) | 2
  Pain in arm or shoulder: Week 93 | 0.00 (0.00)
  Pain in arm or shoulder: Week 96: number analyzed (Participants) | 3
  Pain in arm or shoulder: Week 96 | 0.00 (33.33)
  Pain in arm or shoulder: Week 99: number analyzed (Participants) | 1
  Pain in arm or shoulder: Week 99 | 0.00
  Pain in arm or shoulder: Week 105: number analyzed (Participants) | 1
  Pain in arm or shoulder: Week 105 | 0.00
  Pain in arm or shoulder: Week 111: number analyzed (Participants) | 1
  Pain in arm or shoulder: Week 111 | 0.00
  Pain in arm or shoulder: Week 117: number analyzed (Participants) | 1
  Pain in arm or shoulder: Week 117 | 0.00
  Pain in arm or shoulder: Last visit: number analyzed (Participants) | 73
  Pain in arm or shoulder: Last visit | 0.00 (29.92)
  Pain in other parts: Baseline: number analyzed (Participants) | 75
  Pain in other parts: Baseline | 44.00 (36.42)
  Pain in other parts: Week 6: number analyzed (Participants) | 57
  Pain in other parts: Week 6 | -16.96 (42.78)
  Pain in other parts: Week 9: number analyzed (Participants) | 1
  Pain in other parts: Week 9 | 0.00
  Pain in other parts: Week 12: number analyzed (Participants) | 46
  Pain in other parts: Week 12 | -11.59 (41.70)
  Pain in other parts: Week 15: number analyzed (Participants) | 1
  Pain in other parts: Week 15 | 0.00
  Pain in other parts: Week 18: number analyzed (Participants) | 45
  Pain in other parts: Week 18 | -19.26 (41.74)
  Pain in other parts: Week 21: number analyzed (Participants) | 1
  Pain in other parts: Week 21 | 0.00
  Pain in other parts: Week 24: number analyzed (Participants) | 38
  Pain in other parts: Week 24 | -19.30 (36.87)
  Pain in other parts: Week 27: number analyzed (Participants) | 2
  Pain in other parts: Week 27 | 0.00 (0.00)
  Pain in other parts: Week 30: number analyzed (Participants) | 36
  Pain in other parts: Week 30 | -18.52 (37.75)
  Pain in other parts: Week 33: number analyzed (Participants) | 3
  Pain in other parts: Week 33 | 0.00 (33.33)
  Pain in other parts: Week 36: number analyzed (Participants) | 36
  Pain in other parts: Week 36 | -18.52 (36.90)
  Pain in other parts: Week 39: number analyzed (Participants) | 2
  Pain in other parts: Week 39 | 0.00 (94.28)
  Pain in other parts: Week 42: number analyzed (Participants) | 33
  Pain in other parts: Week 42 | -16.16 (37.38)
  Pain in other parts: Week 45: number analyzed (Participants) | 4
  Pain in other parts: Week 45 | -8.33 (56.93)
  Pain in other parts: Week 48: number analyzed (Participants) | 30
  Pain in other parts: Week 48 | -12.22 (34.45)
  Pain in other parts: Week 51: number analyzed (Participants) | 2
  Pain in other parts: Week 51 | 0.00 (47.14)
  Pain in other parts: Week 54: number analyzed (Participants) | 29
  Pain in other parts: Week 54 | -14.94 (38.41)
  Pain in other parts: Week 57: number analyzed (Participants) | 5
  Pain in other parts: Week 57 | -13.33 (38.01)
  Pain in other parts: Week 60: number analyzed (Participants) | 26
  Pain in other parts: Week 60 | -15.38 (34.29)
  Pain in other parts: Week 63: number analyzed (Participants) | 3
  Pain in other parts: Week 63 | -44.44 (38.49)
  Pain in other parts: Week 66: number analyzed (Participants) | 22
  Pain in other parts: Week 66 | -10.61 (39.02)
  Pain in other parts: Week 69: number analyzed (Participants) | 4
  Pain in other parts: Week 69 | -8.33 (41.94)
  Pain in other parts: Week 72: number analyzed (Participants) | 20
  Pain in other parts: Week 72 | -15.00 (33.29)
  Pain in other parts: Week 75: number analyzed (Participants) | 2
  Pain in other parts: Week 75 | -16.67 (23.57)
  Pain in other parts: Week 78: number analyzed (Participants) | 19
  Pain in other parts: Week 78 | -5.26 (27.81)
  Pain in other parts: Week 81: number analyzed (Participants) | 2
  Pain in other parts: Week 81 | -16.67 (23.57)
  Pain in other parts: Week 84: number analyzed (Participants) | 11
  Pain in other parts: Week 84 | -12.12 (22.47)
  Pain in other parts: Week 87: number analyzed (Participants) | 3
  Pain in other parts: Week 87 | -22.22 (38.49)
  Pain in other parts: Week 90: number analyzed (Participants) | 6
  Pain in other parts: Week 90 | 0.00 (36.51)
  Pain in other parts: Week 93: number analyzed (Participants) | 2
  Pain in other parts: Week 93 | 33.33 (47.14)
  Pain in other parts: Week 96: number analyzed (Participants) | 1
  Pain in other parts: Week 96 | -33.33
  Pain in other parts: Week 99: number analyzed (Participants) | 1
  Pain in other parts: Week 99 | 0.00
  Pain in other parts: Week 105: number analyzed (Participants) | 1
  Pain in other parts: Week 105 | 0.00
  Pain in other parts: Week 111: number analyzed (Participants) | 1
  Pain in other parts: Week 111 | 0.00
  Pain in other parts: Week 117: number analyzed (Participants) | 1
  Pain in other parts: Week 117 | 0.00
  Pain in other parts: Last visit: number analyzed (Participants) | 69
  Pain in other parts: Last visit | -12.56 (37.96)

ADVERSE EVENTS:
Time Frame: Baseline to up to 28 days after the last dose of alectinib (up to 284 weeks)
Description: Safety population
Groups:
- Alectinib 600 mg (Fed): Phase I: Participants received single dose of 20 or 40 or 150 mg alectinib capsules orally to make a dose of 600 mg on Cycle 1 Day -3 and then received 600 mg BID dose for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
- Alectinib 900 mg (Fed): Phase I: Participants received single dose of 20 or 40 or 150 mg alectinib capsules orally to make a dose of 900 mg on Cycle 1 Day -3 and then received 900 mg BID dose for 3-weekly cycles until disease progression, death or withdrawal for any other reasons.
Arm/Group | Alectinib 300 mg (Fasted): Phase I | Alectinib 460 mg (Fed): Phase I | Alectinib 600 mg (Fed): Phase I | Alectinib 760 mg (Fed): Phase I | Alectinib 900 mg (Fed): Phase I | Alectinib 600 mg (Fed): Phase II
All-Cause Mortality (participants affected / at risk) | 7/7 | 4/7 | 6/13 | 2/7 | 9/13 | 45/87
Serious Adverse Events (participants affected / at risk) | 1/7 | 2/7 | 6/13 | 0/7 | 1/13 | 21/87
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 12/13 | 7/7 | 13/13 | 85/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alectinib 300 mg (Fasted): Phase I (N=7) | Alectinib 460 mg (Fed): Phase I (N=7) | Alectinib 600 mg (Fed): Phase I (N=13) | Alectinib 760 mg (Fed): Phase I (N=7) | Alectinib 900 mg (Fed): Phase I (N=13) | Alectinib 600 mg (Fed): Phase II (N=87)
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerebral ventricle dilatation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Stroke-like migraine attacks after radiation therapy (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alectinib 300 mg (Fasted): Phase I (N=7) | Alectinib 460 mg (Fed): Phase I (N=7) | Alectinib 600 mg (Fed): Phase I (N=13) | Alectinib 760 mg (Fed): Phase I (N=7) | Alectinib 900 mg (Fed): Phase I (N=13) | Alectinib 600 mg (Fed): Phase II (N=87)
Fatigue (General disorders) | 4 | 3 | 3 | 5 | 7 | 36
Oedema peripheral (General disorders) | 1 | 1 | 2 | 2 | 3 | 22
Pain (General disorders) | 0 | 0 | 3 | 0 | 1 | 9
Pyrexia (General disorders) | 0 | 1 | 2 | 0 | 0 | 5
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 5
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2 | 3 | 2 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 0 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 5 | 2 | 1 | 12
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 3 | 0 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 0 | 5
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 4 | 1 | 4 | 1 | 20
Alanine aminotransferase increased (Investigations) | 1 | 3 | 3 | 2 | 1 | 16
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 2 | 2 | 1 | 18
Blood bilirubin increased (Investigations) | 0 | 1 | 3 | 1 | 2 | 10
Blood creatinine increased (Investigations) | 0 | 1 | 4 | 1 | 0 | 5
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 1 | 1 | 12
Electrocardiogram PR Prolongation (Investigations) | 0 | 0 | 2 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 1 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 1 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 2 | 0 | 0 | 8
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood phosphorus increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Heart rate irregular (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 6
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 17
Constipation (Gastrointestinal disorders) | 0 | 2 | 3 | 3 | 3 | 34
Nausea (Gastrointestinal disorders) | 2 | 2 | 3 | 0 | 3 | 22
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 3 | 21
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 14
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 5
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 4 | 25
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 1 | 1 | 8
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 1 | 1 | 12
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 5
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Aura (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Narcolepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 3 | 0 | 1 | 14
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 2 | 9
Pneumonia (Infections and infestations) | 0 | 0 | 3 | 0 | 1 | 6
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2 | 3 | 0 | 5
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 3 | 0 | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 3 | 1 | 13
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 1 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 10
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 9
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3 | 0 | 3 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 2 | 1 | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 6
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 0 | 6
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 3 | 0 | 1 | 8
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 1 | 1 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 7
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 1 | 4 | 17
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 6
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 4 | 2 | 0 | 6
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 8
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 1 | 1 | 13
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 7
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 5
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Radiation injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | 2 | 0 | 2 | 7
Flushing (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tanning (Social circumstances) | 0 | 0 | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Babesiosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Blood testosterone decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.